The GlaxoSmithKline group of companies

| Division | ÷ | Worldwide Development |
|------------------|---|-----------------------------------|
| Information Type | : | Reporting and Analysis Plan (RAP) |

| Title | : | Reporting and Analysis Plan (for Group 1 reporting) for a randomized, open-label study to characterize the pharmacokinetics of inhaled oxytocin (GR121619) compared with IM oxytocin in women in the third stage of labour, and with IV oxytocin in non-pregnant, non-lactating women of childbearing potential. |
|---|---|---|
| <b>Compound Number</b> | : | GR121619 |
| <b>Effective Date</b> | : | 08-MAY-2019 |

## **Description:**

- The purpose of this RAP is to describe the planned analyses and output to be included in the Clinical Study Report for Protocol 205920.
- This RAP is intended to describe the Group 1 analyses required for the study.
- This RAP will be provided to the study team members to convey the content of the Statistical Analysis Complete (SAC) deliverable for Group 1.

#### Author(s):

| Author | Date |
|------------------------------------------|------|
| Lead PPD | |
| Senior Statistician (FPD, Biostatistics) | NA |
| Co-Author PPD | INA |
| Statistics Director (FPD, Biostatistics) | |

Copyright 2019 the GlaxoSmithKline group of companies. All rights reserved. Unauthorised copying or use of this information is prohibited.

## The GlaxoSmithKline group of companies

## **RAP Team Review Confirmations (Method: E-mail)**

| Approver | Date |
|---|---|
| Clinical Development Manager, RD PCPS CPSSO | 12-APR-2019 |
| Head, RD Respiratory HUP 2 | 17-APR-2019 |
| Manager, Clinical Pharmacology, CPMS | 15-APR-2019 |
| Manager Data Management, CPSSO Data Management Respiratory 23-APR-2019 | |
| Medical Director, SERM, CMO GCSP SERM US | 12-APR-2019 |
| Principal Programmer/Analyst, RD PCPS Qsci Clinical Statistics 9B2 | 29-APR2019 |

## **Clinical Statistics and Clinical Programming Line Approvals**

## (Method: Pharma TMF eSignature)

| Approver | | Date |
|---|---|---|
| PPD | | |
| Biostatistics and Programming Manager (Infectious Diseases),<br>Biostatistics India | | 08-MAY-2019 |
| On behalf of PPD | (Line Manager, FPD, Biostatistics India) | |
| PPD | | |
| Programming Manager (FPD), RD PCPS Qsci Clinical Statistics 98-MAY-2019 | | |

## **TABLE OF CONTENTS**

| | | | PAGE |
|---|---|---|---|
| 1. | INTRO | ODUCTION | 5 |
| 2. | SLIMI | MARY OF KEY PROTOCOL INFORMATION | 5 |
| ۷. | 2.1. | Changes to the Protocol Defined Statistical Analysis Plan | |
| | 2.1. | Study Objective(s) and Endpoint(s) | 5<br>6 |
| | 2.3. | Study Objective(s) and Endpoint(s) | |
| | 2.4. | Statistical Hypotheses / Statistical Analyses | |
| 3. | DI AN | INED ANALYSES: GROUP 1 | 44 |
| J. | 3.1. | Interim Analyses: Group 1 | |
| | 3.2. | | |
| 4. | ΔΝΔΙ | YSIS POPULATIONS | 12 |
| т. | 4.1. | | |
| 5. | CONS | SIDERATIONS FOR DATA ANALYSES AND DATA HANDLING | |
| | | VENTIONS | 13 |
| | 5.1. | Study Treatment & Sub-group Display Descriptors: Group 1 | |
| | 5.2. | Baseline Definitions | |
| | 5.3. | Other Considerations for Data Analyses and Data Handling Conventions | 14 |
| 6. | CTLID | DY POPULATION ANALYSES: GROUP 1 | 15 |
| 0. | 6.1. | Overview of Planned Study Population Analyses | |
| 7. | 0455 | | |
| 1. | 7.1. | TY ANALYSES: GROUP 1Adverse Events Analyses | |
| | 7.1.<br>7.2. | • | |
| | 7.2.<br>7.3. | Clinical Laboratory Analyses | |
| | | Other Safety Analyses | |
| 8. | | RMACOKINETIC ANALYSES : GROUP 1 | |
| | 8.1. | Primary Pharmacokinetic Analyses : Group 1 | |
| | | 8.1.1. Endpoint / Variables : Group 1 | |
| | | 8.1.1.1. Drug Concentration Measures : Group 1 | |
| | | 8.1.1.2. Derived Pharmacokinetic Parameters: Group 1 | |
| | | 8.1.2. Summary Measure: Group 1 | |
| | | 8.1.3. Population of Interest: Group 1 | |
| | 8.2. | POPULATION PHARMACOKINETIC (POPPK) ANALYSES | |
| | 8.3. | Secondary Pharmacokinetic Analyses: Group 1 | |
| | 0.4 | 8.3.1. Endpoint / Variables : Group 1 | |
| | 8.4. | Exploratory Pharmacodynamic Analyses: Group 1 | |
| | | 8.4.1. Endpoint / Variables: Group 1 | |
| | | 8.4.2. Summary Measure: Group 1 | |
| | | 8.4.3. Population of Interest: Group 1 | 19 |
| 9. | REFE | ERENCES | 20 |
| 10 | ∆ DD⊏ | INDICES | 21 |

| 10.1. | | x 1: Protocol Deviation Management and Definitions for Per Population | 21 |
|---|---|---|---|
| 10.2. | | x 2: Schedule of Activities | |
| 10.2. | 10.2.1. | Protocol Defined Schedule of Events : Group 1 | |
| | 10.2.1. | 10.2.1.1. Time & Events General Overview | |
| | | 10.2.1.2. Time & Events General Overview | |
| 10.3. | Annondi | x 3: Assessment Windows | |
| 10.3. | | x 4: Study Phases and Treatment Emergent Adverse | 24 |
| 10.4. | | 4. Study Friases and Treatment Emergent Adverse | 25 |
| | 10.4.1. | | |
| | | 10.4.1.1. Study Phases for Concomitant Medication | |
| | 10.4.2. | Treatment Emergent Flag for Adverse Events | |
| 10.5. | | x 5: Data Display Standards & Handling Conventions | |
| | 10.5.1. | Reporting Process | |
| | 10.5.2. | Reporting Standards | |
| | 10.5.3. | Reporting Standards for Pharmacokinetic | |
| 10.6. | Appendix | x 6: Derived and Transformed Data | |
| | 10.6.1. | General | |
| | 10.6.2. | Study Population | |
| | 10.6.3 | Safety | |
| 10.7. | Appendix | x 7: Reporting Standards for Missing Data | 32 |
| | 10.7.1. | | |
| | 10.7.2. | Handling of Missing Data | |
| | | 10.7.2.1. Handling of Missing and Partial Dates | 32 |
| 10.8. | Appendix | x 8: Values of Potential Clinical Importance | |
| | | Laboratory Values | |
| | 10.8.2. | Vital Signs | 34 |
| 10.9. | | x 9: Abbreviations & Trade Marks | |
| | 10.9.1. | Abbreviations | 35 |
| | 10.9.2. | Trademarks | 36 |
| 10.10. | Appendix | x 10: List of Data Displays | 37 |
| | | Data Display Numbering | |
| | 10.10.2. | Mock Example Shell Referencing | 37 |
| | 10.10.3. | Deliverables | 37 |
| | 10.10.4. | Study Population Tables | 38 |
| | 10.10.5. | Pharmacokinetic Tables | 39 |
| | | Pharmacokinetic Figures | |
| | 10.10.7. | Safety Tables | 41 |
| | 10.10.8. | Safety Figure | 43 |
| | 10.10.9. | ICH Listings | 44 |
| | | .Non-ICH Listings | |
| 10.11. | Appendix | x 11: Mock Shell | 46 |

## 1. INTRODUCTION

The purpose of this reporting and analysis plan (RAP) is to describe the analyses of Group 1 to be included in the Clinical Study Report for Protocol:

| Revision Chronology: | | |
|---|---|---|
| 2016N281575_00 | 2016-AUG-22 | Original |
| 2016N281575_01 | 2016-OCT-10 | Section 6.2: Inclusion of information on CE marking. |
| 2016N281575_02 | 2018-JAN-04 | Update to PK collection procedures and implementation of instream PK data analysis. |
| | | Update to location of Secondary Medical Monitor contact information. |
| 2016N281575_03 | 2018-MAY-30 | Modification to informal interim and Group 2 analysis plans. |

## 2. SUMMARY OF KEY PROTOCOL INFORMATION

## 2.1. Changes to the Protocol Defined Statistical Analysis Plan

Changes from the originally planned statistical analysis specified in the protocol are outlined in Table 1.

Table 1 Changes to Protocol Defined Analysis Plan

| Protocol | Reporting & Analysis Plan | |
|---|---|---|
| Statistical Analysis Plan | Statistical Analysis Plan | Rationale for Changes |
| To compare pharmacokinetics of<br>IH oxytocin to 10 I.U. IM<br>oxytocin in women in TSL. | To produce summary<br>statistics for IH and IM<br>Oxytocin | Due to sparse PK concentration available for IM and IH Oxytocin a formal statistical analysis comparison is not possible; summary statistics will be presented instead. |
| To characterize the pharmacokinetics of single doses of IH oxytocin and 10 International Units (I.U.) IM oxytocin in women in TSL. | To produce individual plasma concentration-time plots and summary statistics for PK parameters: Maximum observed plasma concentration (Cmax), Observed plasma concentrations at 10 minutes (min) postdose (Cp10), Observed plasma concentrations at 20 min post-dose (Cp20), Observed plasma concentrations at 30 min post-dose (Cp30), Time to Cmax (tmax), Area under | As only sparse PK concentration is available for IM and IH Oxytocin PK parameters will be derived wherever data permit. Terminal Phase half-life (t1/2) will not be calculated. AUC(0-3h) will not be calculated instead AUC(0-t) and time of last quantifiable concentration will be computed. |

| Protocol | Reporting & Analysis Plan | |
|---|---|---|
| Statistical Analysis Plan | Statistical Analysis Plan | Rationale for Changes |
| | concentration-time curve from time zero to the time of the last quantifiable concentration (AUC(0-t)),as data permit. Terminal Phase half-life (t1/2) will not be calculated | |
| To compare pharmacokinetics of<br>IH oxytocin between Group 1<br>and Group 2 | No statistical comparison<br>will be done | As only sparse PK concentration is available for IH Oxytocin in Group 1 as compared to Group 2, a statistical comparison will not be reported. |
| All Subjects Population | All Subjects population label changed to Safety population. | To be compliant with the<br>new RAP template |
| Enrolled Population (Defined as all subjects who were enrolled for the trial irrespective of whether they were randomized or not and for whom a record exists on the study database. This population will be used for summarizing screening failure reasons. | All participants who passed screening and entered the study including randomized participants and run in failures Note: Screening failures (who never passed screening even if rescreened) and participants screened but never enrolled into the study (Reserve, Not Used) are excluded from the Enrolled population as they did not enter the study. | To be compliant with the new RAP template |

# 2.2. Study Objective(s) and Endpoint(s)

Group 1 – Women in Third Stage of Labour (TSL)op

| Objectives | Endpoints |
|---|---|
| Primary Objectives | Primary Endpoints |
| To characterize the pharmacokinetics<br>of single doses of IH oxytocin and 10<br>International Units (I.U.) IM oxytocin in<br>women in TSL. | <ul> <li>Plasma concentration time profile for IH oxytocin and 10 I.U. IM oxytocin.</li> <li>PK parameters: Maximum observed plasma concentration (Cmax), Observed plasma concentrations at 10 minutes (min) postdose (Cp10), Observed plasma concentrations at 20 min post-dose (Cp20), Observed plasma concentrations at 30 min post-dose (Cp30), Time to Cmax (tmax), Area under concentration-time curve (AUC), and Terminal phase half-life (t1/2) will be calculated as data permit.</li> </ul> |
| Secondary Objectives | Secondary Endpoints |
| <ul> <li>To evaluate the safety and tolerability<br/>of inhaled oxytocin.</li> </ul> | General safety parameters: adverse events (AE); absolute values and changes over time of vital signs (blood pressure, heart rate, respiratory rate, temperature). |

| Objectives | Endpoints |
|---|---|
| To compare pharmacokinetics of IH oxytocin to 10 I.U. IM oxytocin in women in TSL. | Cmax, Cp10, Cp20, Cp30, Area under the concentration-<br>time curve from time zero (pre-dose) to three hours (h)<br>(AUC[0-3h]) will be compared as data permit. |
| Exploratory Objectives | Exploratory Endpoints |
| Pharmacodynamic effect of IH<br>oxytocin and 10 I.U. IM oxytocin in<br>women in TSL. | Pre and post-delivery haemoglobin |
| Participant feedback regarding ease of use, instructions, and perceived ability of patients to use the ROTAHALER. | Questionnaire results from participants. |

Group 2 - Non-pregnant, non-lactating females of child bearing potential

| Obj | ectives | End | points |
|---|---|---|---|
| Prin | mary Objectives | Prin | nary Endpoints |
| • | To evaluate the safety and tolerability of IH and IV Oxytocin | | General safety parameters: adverse events; absolute values and changes over time of vital signs (blood pressure, heart rate) and 12-lead electrocardiogram (ECG) parameters (PR, QRS, QT, Corrected QT interval [QTc] intervals) from pre-dose values. Specific respiratory safety parameters: adverse respiratory events as monitored by spirometry including Forced expiratory volume at 1 minute (FEV1.0), respiratory rate, and pulse oximetry. |
| • | To characterize the pharmacokinetics of single doses of IH oxytocin and 5 I.U. IV oxytocin. | • | Plasma concentration time profile for IH oxytocin and 5 I.U. IV oxytocin. PK parameters: Cmax, Cp10, Cp20, Cp30, tmax, AUC, Plasma clearance (CL), volume of distribution and t1/2 will be calculated as data permit. |
| Exploratory Objectives | | Exploratory Endpoints | |
| • | To evaluate endogenous plasma oxytocin concentrations in non-pregnant females in the presence and absence of the combined oral contraceptive. | • | Pre-dose plasma concentrations of oxytocin. |
| • | To compare the IH pharmacokinetics of oxytocin between Cohort A (subjects on combined oral contraceptive) and Cohort B (subjects using a non-hormonal form of contraception). | • | Cp10, Cp20, Cp30, Cmax, AUC(0-3h), Area under the concentration time curve from time zero to infinity (AUC[0-∞]) and t1/2, will be compared as data permit. |
| • | To compare the IV pharmacokinetics of oxytocin between Cohort A and Cohort B. | | Cmax, AUC, t1/2, CL and Volume of distribution (VOD) will be compared as data permit. |

## Groups 1 and 2 – Women in TSL and Non-pregnant, non-lactating females of child bearing potential

| Objectives | Endpoints |
|---|---|
| Primary Objectives | Primary Endpoints |
| To compare pharmacokinetics of IH oxytocin between Group 1 and Group 2 | <ul> <li>Cp10, Cp20, Cp30, Cmax, AUC(0-3h) AUC(0-∞), and<br/>t1/2 will be compared as data permit.</li> </ul> |

### 2.3. Study Design



| Overview of St | Overview of Study Design and Key Features |
|---|---|
| | of two dosing sessions: C: 400 mcg IH oxytocin D: 5 I.U. IV oxytocin |
| Interim<br>Analysis | <ul> <li>No formal Interim Analysis are planned, however, PK samples will be analysed and<br/>preliminary PK parameters derived following completion of approximately 5 women on<br/>each treatment group: 400 mcg IH and 10 I.U. IM to women in TSL (Group 1) and 400<br/>mcg IH to non-pregnant women on the combined oral contraceptive (Group 2 Cohort<br/>A), in order to assess if dose escalation is required.</li> </ul> |

## 2.4. Statistical Hypotheses / Statistical Analyses

No formal hypotheses will be tested.

For IH and IM oxytocin, summary statistics will be produced separately for IH Oxytocin and IM Oxytocin. Due to sparse PK concentrations, it is not possible to include a formal statistical analysis to compare IH and IM Oxytocin. PK parameters will be derived as data permit. Individual plots, listings and summary tables will be produced for available PK concentration data. Only listings and summary tables will be produced for PK Parameter data.

#### 3. PLANNED ANALYSES: GROUP 1

## 3.1. Interim Analyses: Group 1

No formal Interim Analysis are planned, however, PK samples will be analysed and preliminary PK parameters derived following completion of approximately 5 women on each treatment group: 400 mcg IH and 10 I.U. IM to women in TSL (Group 1) and 400 mcg IH to non-pregnant women on the combined oral contraceptive (Group 2 Cohort A), in order to assess if dose escalation is required.

Due to sparse PK concentration-time data available following administration of IH and IM oxytocin to women in TSL, only concentration time plots were presented at the interim analysis. The Study has been terminated early due the unanticipated inability to be able to quantify plasma oxytocin using a selective and sensitive (LLQ 2pg/mL) analytical assay due to low oxytocin concentrations (<2pg/mL) in the majority of samples collected from women in Third Stage Labour (TSL), following either IM or IH administration. Therefore, the Primary objective of the study to characterise the PK of single doses of IH and IM oxytocin in women in TSL, cannot be met, and the study is being terminated

## 3.2. Final Analyses

The final planned primary analyses for Group 1 will be performed after the completion of the following sequential steps:

- 1. All participants who had enrolled into the study prior to the termination of the study as defined in the protocol will be part of final analysis.
- 2. All required database cleaning activities have been completed for group 1 and final database release (DBR) and database freeze (DBF) for group 1 has been declared by Data Management.
- 3. All criteria for unblinding the randomization codes for group 1 have been met.
- 4. Randomization codes for group 1 have been distributed according to RandAll NG procedures.

#### 4. ANALYSIS POPULATIONS

| Population | Definition / Criteria | Analyses Evaluated |
|---|---|---|
| Screened | All participants who were screened for eligibility | <ul> <li>Screen Failures</li> </ul> |
| Enrolled | All participants who passed screening and entered the study including randomized participants and run in failures Note: Screening failures (who never passed screening even if rescreened) and participants screened but never enrolled into the study (Reserve, Not Used) are excluded from the Enrolled population as they did not enter the study. | Study Population |
| Safety | Comprise of subjects who receive at least one dose of study medication. This population will be used for the study population and safety displays. Note: This population will be based on the treatment the participants actually received | <ul><li>Study Population</li><li>Safety</li></ul> |
| Pharmacokinetic<br>(PK) | Subjects in the 'Safety' population for whom a pharmacokinetic sample was obtained and analysed. PK population will be the population for reporting PK data. | • PK |

Refer to Appendix 10: List of Data Displays which details the population used for each display.

#### 4.1. Protocol Deviations

Protocol deviations will be tracked by the study team throughout the conduct of the study in accordance with the Protocol Deviation Management Plan.

- o Data will be reviewed prior to freezing the database to ensure all important deviations are captured and categorised on the protocol deviations dataset.
- o The SI dataset will include all protocol deviations; the analysis dataset will include only important protocol deviations. The analysis dataset will be used for the listing of important protocol deviations.
- The study endpoints will be reported using the populations detailed in Section 4 of this document regardless of whether the participants deviate from the protocol.
- A separate listing of all inclusion/exclusion criteria deviations will also be provided. This listing will be based on data as recorded on the inclusion/exclusion page of the eCRF.

# 5. CONSIDERATIONS FOR DATA ANALYSES AND DATA HANDLING CONVENTIONS

## 5.1. Study Treatment & Sub-group Display Descriptors: Group 1

| Treatment Group Descriptions | | | |
|---|---|---|---|
| RandAll NG Data Displays for Reporting | | | |
| Code | Description | Description | Order in TLF |
| А | 400 mcg IH oxytocin | 400 mcg IH | 1 |
| В | 10 I.U. IM oxytocin | 17 mcg IM | 2 |

The treatment dosage will be included in the footnotes for the respective tables/listings. If treatment codes have been displayed in the tables/listings the treatment descriptions should be included as footnotes.

#### 5.2. Baseline Definitions

For all endpoints (except as noted in baseline definitions) the baseline value will be the latest pre-dose assessment with a non-missing value. If time is not collected, Day 1 assessments are assumed to be taken prior to first dose and used as baseline. Unscheduled visits will not be used for baseline calculation

Baseline definitions for Group 1

| Parameter | Study Asses | Baseline Used in<br>Data Display | | |
|---|---|---|---|---|
| | Screening | | | |
| Safety | | | | |
| Vital Signs (blood pressure, heart rate, temperature, respiratory rate) | Х | Х | X | Day 1 |
| LAB | Х | | | Screening |

Unless otherwise stated, if baseline data is missing no derivation will be performed and baseline will be set to missing.

# 5.3. Other Considerations for Data Analyses and Data Handling Conventions

Other considerations for data analyses and data handling conventions are outlined in the appendices:

| Section | Component |
|---------|----------------------------------------------------------------|
| 10.3 | Appendix 3: Assessment Windows |
| 10.4 | Appendix 4: Study Phases and Treatment Emergent Adverse Events |
| 10.5 | Appendix 5: Data Display Standards & Handling Conventions |
| 10.6 | Appendix 6: Derived and Transformed Data |
| 10.7 | Appendix 7: Reporting Standards for Missing Data |
| 10.8 | Appendix 8: Values of Potential Clinical Importance |

## 6. STUDY POPULATION ANALYSES: GROUP 1

## 6.1. Overview of Planned Study Population Analyses

The study population analyses will be based on the Safety & Enrolled population, with screen failures as an exception.

Study population analyses including analyses of subject's disposition, protocol deviations, demographic and baseline characteristics, prior and concomitant medications, and exposure and treatment compliance will be based on GSK Core Data Standards.

Details of the planned displays are provided in Appendix 10: List of Data Displays and will be based on GSK data standards and statistical principles.

#### 7. SAFETY ANALYSES: GROUP 1

The safety analyses will be based on the Safety population, unless otherwise specified.

## 7.1. Adverse Events Analyses

Adverse events analyses including the analysis of adverse events (AEs), Serious (SAEs) and other significant AEs will be based on GSK Core Data Standards. The details of the planned displays are provided in Appendix 10: List of Data Displays.

## 7.2. Clinical Laboratory Analyses

Laboratory evaluations including the analyses of Chemistry laboratory tests, Hematology laboratory tests, Urinalysis, and liver function tests will be based on GSK Core Data Standards. The details of the planned displays are in Appendix 10: List of Data Displays.

## 7.3. Other Safety Analyses

The analyses of non-laboratory safety test results including ECGs and vital signs will be based on GSK Core Data Standards, unless otherwise specified. The details of the planned displays are presented in Appendix 10: List of Data Displays.

## 8. PHARMACOKINETIC ANALYSES: GROUP 1

### 8.1. Primary Pharmacokinetic Analyses: Group 1

#### 8.1.1. Endpoint / Variables : Group 1

- Plasma concentration time profile for IH oxytocin and 10 I.U. IM oxytocin.
- PK parameters: Maximum observed plasma concentration (Cmax), Observed plasma concentrations at 10 minutes (min) postdose (Cp10), Observed plasma concentrations at 20 min post-dose (Cp20), Observed plasma concentrations at 30 min post-dose (Cp30), Time to Cmax (tmax), Area under concentration-time curve (AUC(0-t)), and time of last quantifiable concentration will be calculated as data permit.

#### 8.1.1.1. Drug Concentration Measures : Group 1

Refer to Appendix 5: Data Display Standards & Handling Conventions (Section 10.5.2 and Section 10.5.3 Reporting Standards for Pharmacokinetic)

#### 8.1.1.2. Derived Pharmacokinetic Parameters: Group 1

Pharmacokinetic parameters will be calculated by standard non-compartmental analysis according to current working practices and GSK procedures using the currently supported version of WinNonlin. All calculations of non-compartmental parameters will be based on actual sampling times. Pharmacokinetic parameters listed will be determined from the plasma concentration-time data, as data permits.

| Treatment | Parameter | Parameter Description |
|---|---|---|
| IH/IM | Cmax | Maximum observed concentration, determined directly from the concentration-time data. |
| IH/IM | Cp10 | Quantified concentration in PK sample collected at 10 minutes (nominal time) post-dose, determined directly from the concentration-time data. |
| IH/IM | Cp20 | Quantified concentration in PK sample collected at 20 minutes (nominal time) post-dose, determined directly from the concentration-time data. |
| IH/IM | Cp30 | Quantified concentration in PK sample collected at 30 minutes (nominal time) post-dose, determined directly from the concentration-time data. |
| IH/IM | tmax | Time to reach Cmax, determined directly from the concentration-time data. |
| IH/IM | AUC(0-t) | Area under the concentration-time curve from time zero to the time of the last quantifiable concentration (C(t)) will be calculated using the linear trapezoidal rule for each incremental trapezoid and the log trapezoidal rule for each decremental trapezoid. |
| IH/IM | tlast | Time of last quantifiable concentration |

At least 2 quantifiable (3 including time 0 where NQ values at time zero will be set to 0) values per profile are required to calculate the AUC(0-t). For profiles with less than 2 quantifiable values, AUC(0-t) will be coded with NC in the PKPar file.

#### 8.1.2. Summary Measure: Group 1

Pharmacokinetic concentration data will be presented in graphical and/or tabular form and will be summarized descriptively by IH oxytocin and IM Oxytocin.

The conversion factor to normalise IM doses is 1 IU = 1.7 mcg oxytocin

As a large number of PK parameter values will be reported as Non Calculable (NC: PK parameter cannot be derived due to the presence of non-quantifiable data) then the PK parameter will be summarised by following measures

- number of subjects with non-missing observations, n, (includes those reported as NC)
- number of subjects for whom parameter cannot be derived because of NQ concentrations, n\*, (reported as NC)
  - median, minimum and maximum

In addition a frequency table of the number of subjects with all concentrations NQ and the number of subjects with one, or 2 or more measurable concentrations will be produced.

#### 8.1.3. Population of Interest: Group 1

The primary pharmacokinetic analyses will be based on the Pharmacokinetic population, unless otherwise specified.

# 8.2. POPULATION PHARMACOKINETIC (POPPK) ANALYSES

PK samples will be analysed periodically throughout the study duration to enable development of a preliminary population PK model. If appropriate, a population PK analysis may also be conducted on the final data. In addition the oxytocin plasma concentration-time data may be merged with historical data and analysed as part of a population PK meta-analysis. The timeline for these analyses will be independent of the analysis described in this RAP. To support this analysis a NONMEM-specific data file will be generated, the specifications of which are provided in POP PK RAP appendix.

## 8.3. Secondary Pharmacokinetic Analyses: Group 1

#### 8.3.1. Endpoint / Variables : Group 1

• Cmax, Cp10, Cp20, Cp30, Area under the concentration-time curve from time zero (pre-dose) to three hours (h) (AUC[0-3h]) will be compared as data permit.

Due to sparse PK concentrations, it is not possible to include a formal statistical analysis to compare IH and IM Oxytocin therefore no statistical analysis will be performed.

## 8.4. Exploratory Pharmacodynamic Analyses: Group 1

### 8.4.1. Endpoint / Variables: Group 1

- Pre and post-delivery haemoglobin
- Questionnaire results from participants

### 8.4.2. Summary Measure: Group 1

Pre and post-delivery Haemoglobin will be summarized and listed along with other haematology parameters. A box plot will be produced for pre and post-delivery haemoglobin.

A listing and a summary table will be produced for the questionnaire results from the Rotahaler.

## 8.4.3. Population of Interest: Group 1

The exploratory analyses will be based on the Safety population, unless otherwise specified.

## 9. REFERENCES

GlaxoSmithKline Document Number 2016N281575\_03: A randomized, open-label study to characterize the pharmacokinetics of IH oxytocin (GR121619) compared with IM oxytocin in women in the third stage of labour, and with IV oxytocin in non-pregnant, non-lactating women of childbearing potential. (amendment no.3 – 30-May-2018)

## 10. APPENDICES

# 10.1. Appendix 1: Protocol Deviation Management and Definitions for Per Protocol Population

This section is not applicable as Per Protocol Population is not defined for this study.

## 10.2. Appendix 2: Schedule of Activities

### 10.2.1. Protocol Defined Schedule of Events: Group 1

### 10.2.1.1. Time & Events General Overview

## Group 1

| | 8 | | Study Day | 11000-1100 |
|---|---|---|---|---|
| Procedure | Screening <sup>4</sup> | Main Phase | Follow – Up 1 (approx. 24 hours post dose) | Follow – Up 2 (7-14 days post dose) |
| Informed Consent and Demography | X | | 1 2 | |
| Brief Physical Examination | Х | | | |
| Medical history (incl. substance abuse) | Х | | | |
| Inhaler device training / education session | X | | | |
| Laboratory assessments <sup>1</sup> | X | | | |
| Vital signs <sup>2</sup> | Х | χ | | |
| Pharmacokinetic blood sample | " | χ | | |
| Oxytocin Administration (IM/IH) | 2 | Χ | | |
| Full blood count | | χ | | |
| Labour Events Documentation | | Χ | | |
| Device acceptability questionnaire3 | | Χ | | |
| Prior / concomitant medication review | X | Χ | X | Χ |
| AE review | | | continuous review | |
| SAE review | continuous review | | | |

- 1. Only required if done as part of routine care. Additional study-specific laboratory assessments not required.
- 2. Includes blood pressure, heart rate, temperature, respiratory rate
- 3. Only to be used when randomized to IH oxytocin
- 4. To be completed after 18th week of pregnancy (based on estimated date of delivery).

#### 10.2.1.2. Time & Events - Main Phase Procedures

## Group 1

| | | | Time post dose | | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Procedure | Pre- | 3 min | 5 min | 10 | 15 min | 20 | 30 | 1 hr | 2 hr | 2.5 hr | 3 hr | 4 hr |
| | dose | | | min | | min | min | | | | | |
| Vital signs <sup>1</sup> | | | | | | | χ | | Χ | | | |
| Pharmacokinetic blood sample | χ2 | χ | χ | Χ | χ | Χ | χ | χ | Χ | χ | X | χ |
| Prior medication review | Х | | | | | | | | | | | |
| Concomitant medication review | | | | | | | C( | ontinuous | review | | | |
| AE review | | continuous review | | | | | | | | | | |
| SAE Review | | | | | | 00 | ontinuous | review | | | | |
| Device Acceptability Questionnaire <sup>3</sup> | | | | | | | | | | | | χ |
| Full Blood Count X | | | | | | | | | | | | Х |

- 1. Includes blood pressure, heart rate, temperature, respiratory rate
- 2. Predose PK sample to be taken immediately prior to administration of study treatment
- 3. Only to be administered when randomized to IH oxytocin

## 10.3. Appendix 3: Assessment Windows

No assessment windows will be applied.

# 10.4. Appendix 4: Study Phases and Treatment Emergent Adverse Events

## 10.4.1. Study Phases

Assessments and events will be classified according to the time of occurrence relative to study treatment.

| Study Phase | Definition |
|---|---|
| Pre-Treatment | Date < Study Treatment Start Date |
| On-Treatment | Study Treatment Start Date ≤ Date ≤ Study Treatment Stop Date +1 |
| Post-Treatment | Date > Study Treatment Stop Date +1 |

### 10.4.1.1. Study Phases for Concomitant Medication

| Study Phase | Definition |
|---|---|
| Prior | If medication end date is not missing and is prior to 18th week of pregnancy. |
| Concomitant | Any medication that is not a prior |

#### NOTES:

 Please refer to Appendix 7: Reporting Standards for Missing Data for handling of missing and partial dates for concomitant medication. Use the rules in this table if concomitant medication date is completely missing.

## 10.4.2. Treatment Emergent Flag for Adverse Events

| Flag | Definition |
|---|---|
| Treatment<br>Emergent | If AE onset date is on or after treatment start date & on or before treatment stop date. |
| | • Study Treatment Start Date ≤ AE Start Date ≤ Study Treatment Stop Date +1. |

#### NOTES:

- If the study treatment stop date is missing, then the AE will be considered to be On-Treatment.
- Time of study treatment dosing and start/stop time of AEs should be considered, if collected.

# 10.5. Appendix 5: Data Display Standards & Handling Conventions

#### 10.5.1. Reporting Process

| Software | |
|---|---|
| The currently supported versions of SAS software 9.4 will be used. | |
| Reporting Area | |
| HARP Server | : UK1SALX00175 |
| HARP Compound (Group 1 Dry Run) | : /arenv/arprod/gr121619/mid205920/final_03 |
| HARP Compound (Group 1 Final) /arenv/arprod/gr121619/mid205920/final_04 | |
| Analysis Datasets | |
| Analysis datasets will be created according to Legacy GSK A&R dataset | |
| Generation of RTF Files | |
| RTF files will be generated for summary tables | |

#### 10.5.2. Reporting Standards

#### General

- The current GSK Integrated Data Standards Library (IDSL) will be applied for reporting, unless otherwise stated (IDSL Standards Location: https://spope.gsk.com/sites/IDSLLibrary/SitePages/Home.aspx):
  - 4.03 to 4.23: General Principles
  - 5.01 to 5.08: Principles Related to Data Listings
  - 6.01 to 6.11: Principles Related to Summary Tables
  - 7.01 to 7.13: Principles Related to Graphics

#### **Formats**

- All data will be reported according to the actual treatment the subject received unless otherwise stated.
- GSK IDSL Statistical Principles (5.03 & 6.06.3) for decimal places (DP's) will be adopted for reporting of data based on the raw data collected, unless otherwise stated.
- Numeric data will be reported at the precision collected on the eCRF.
- The reported precision from non eCRF sources will follow the IDSL statistical principles but may be adjusted to a clinically interpretable number of DP's.

#### **Planned and Actual Time**

- Reporting for tables, figures and formal statistical analyses:
  - Planned time relative to dosing will be used in figures, summaries, statistical analyses and calculation of any derived parameters, unless otherwise stated.
  - The impact of any major deviation from the planned assessment times and/or scheduled visit days
    on the analyses and interpretation of the results will be assessed as appropriate.
- Reporting for Data Listings:
  - Planned and actual time relative to study drug dosing will be shown in listings (Refer to IDSL Statistical Principle 5.05.1).
  - Unscheduled or unplanned readings will be presented within the subject's listings.

#### **Unscheduled Visits**

- Unscheduled visits will not be included in summary tables and/or figures.
- All unscheduled visits will be included in listings.

| Descriptive Summary Statistics | |
|---|---|
| Continuous Data | Refer to IDSL Statistical Principle 6.06.1 |
| Categorical Data | N, n, frequency, % |
| Reporting of Pharmac | cokinetic Concentration Data |
| Descriptive Summary | Refer to IDSL Statistical Principle 6.06.1 |
| Statistics | Assign zero to NQ values (Refer to GUI_51487 for further details) |
| Reporting of Pharmac | cokinetic Parameters |
| Summary table | Summary table will be produced as described in Section 8.1.2 |
| Listing | All PK Parameters that are collected will be listed |
| Reporting of No treatment | |
| If in a situation where a subject has received no treatment, then the subject will be included only in Screened and enrolled population. | |
| Graphical Displays | |
| Refer to IDSL Statistical Principals 7.01 to 7.13. | |
| All figures will use coloured lines | |

# 10.5.3. Reporting Standards for Pharmacokinetic

| Pharmacokinetic Concentration Data | |
|---|---|
| PC Windows Non- | WNL file will be produced for PK parameters. |
| Linear (WNL) File | Note: Concentration values will be imputed as per GUI_51487 |
| Descriptive Summary | Refer to IDSL PK Display Standards. |
| Statistics, Graphical | Refer to IDSL Statistical Principle 6.06.1. |
| Displays and Listings | Note: Concentration values will be imputed as per GUI_51487 for descriptive summary statistics/analysis and summarized graphical displays only. |
| NONMEM/Pop PK<br>File | Pop-PK file (CSV format) for the POP-PK analysis by Clinical Pharmacology Modelling and Simulation function will be created according to the data specification detailed in Section 9.1 Data Specification of the Pop-PK RAP (RAP-IVF116828-201558-205920-PopPK, located in Cabinets/Study File/GR121619/_Project/Meta Analysis/ RAP-IVF116828-201558-205920-PopPK) |
| Pharmacokinetic Parameter Derivation | |
| PK Parameter to be | The following PK parameters will be derived by the Programmer: Cp10, Cp20 and |
| Derived by | Cp30 |
| Programmer | |

### 10.6. Appendix 6: Derived and Transformed Data

#### 10.6.1. General

#### **Multiple Measurements at One Analysis Time Point**

- Mean of the measurements will be calculated and used in any derivation of summary statistics but if listed, all data will be presented.
- Participants having both High and Low values for Normal Ranges at any post-baseline visit for safety parameters will be counted in both the High and Low categories of "Any visit post-baseline" row of related summary tables. This will also be applicable to relevant Potential Clinical Importance summary tables.

#### **Study Day**

- Calculated as the number of days from First Dose Date:
  - Ref Date = Missing → Study Day = Missing
  - Ref Date < First Dose Date → Study Day = Ref Date First Dose Date
  - Ref Data ≥ First Dose Date → Study Day = Ref Date (First Dose Date) + 1

## 10.6.2. Study Population

#### **Demographics**

#### Age

- GSK standard IDSL algorithms will be used for calculating age.
- Randomization date will be used as reference date to calculate age

#### **Body Mass Index (BMI)**

Calculated as Weight (kg) / [Height (m)<sup>2</sup>

#### **Extent of Exposure**

Number of days of exposure to study drug will be calculated based on the formula:

#### Duration of Exposure in Days = Treatment Stop Date - (Treatment Start Date) + 1

Participants who were randomized but did not report a treatment start date will be categorised as
having zero days of exposure. If there are any treatment breaks during the study, exposure data will be
adjusted accordingly.

## 10.6.3 Safety

#### **ECG Parameters**

#### RR Interval

• IF RR interval (msec) is not provided directly, then RR can be derived as :

[1] If QTcB is machine read & QTcF is not provided, then:

$$RR = [(QT/QTcB)^{2}]^{1000}$$

[2] If QTcF is machine read and QTcB is not provided, then:

$$RR = [(QT/QTcF)^{3}]^{1000}$$

• If ECGs are manually read, the RR value preceding the measurement QT interval should be collected values THEN do not derive.

#### **Corrected QT Intervals**

- When not entered directly in the eCRF, corrected QT intervals using Bazett's (QTcB) and Fredericia's (QTcF) formulas will be calculated, in msec, depending on the availability of other measurements.
- IF RR interval (msec) is provided or calculated then missing QTcB and/or QTcF will be derived as :

$$QTcB = \frac{QT}{\sqrt{\frac{RR}{1000}}}$$

$$QTcF = \frac{QT}{3\sqrt{\frac{RR}{1000}}}$$

#### **Laboratory Parameters**

- If a laboratory value which is expected to have a numeric value for summary purposes, has a non-detectable level reported in the database, where the numeric value is missing, but typically a character value starting with '<x' or '>x' (or indicated as less than x or greater than x in the comment field) is present, the number of significant digits in the observed values will be used to determine how much to add or subtract in order to impute the corresponding numeric value.
  - Example 1: 2 Decimal Points = '< x' becomes x 0.01
  - Example 2: 1 Decimal Point = '> x' becomes x + 0.1
  - Example 3: 0 Decimal Points = '< x' becomes x 1</p>

## 10.7. Appendix 7: Reporting Standards for Missing Data

## 10.7.1. Premature Withdrawals

| Element | Reporting Detail |
|---|---|
| General | <ul> <li>Subject study completion (i.e. as specified in the protocol) was defined as who has completed all phases of the study including the follow-up visit(s).</li> <li>Withdrawn subjects may be replaced in the study.</li> <li>All available data from participants who were withdrawn from the study will be listed and all available planned data will be included in summary tables and figures, unless otherwise specified.</li> </ul> |

## 10.7.2. Handling of Missing Data

| Element | Reporting Detail |
|---|---|
| General | Missing data occurs when any requested data is not provided, leading to blank fields on the collection instrument: |
| | <ul> <li>These data will be indicated by the use of a "blank" in subject listing displays.</li> <li>Unless all data for a specific visit are missing in which case the data is excluded from the table.</li> </ul> |
| | <ul> <li>Answers such as "Not applicable" and "Not evaluable" are not considered to be<br/>missing data and should be displayed as such.</li> </ul> |
| Outliers | Any participants excluded from the summaries and/or statistical analyses will be documented along with the reason for exclusion in the clinical study report. |

## 10.7.2.1. Handling of Missing and Partial Dates

| Element | Reporting Detail |
|---|---|
| General | Partial dates will be displayed as captured in subject listing displays. |
| Adverse Events | <ul> <li>The eCRF does not allow for the possibility of partial dates. The eCRF and the site need to enter the full date or if not known, they would be required to complete an item level comment bubble to specify why the date is unknown. This would also be documented in the Data Quality Release Report by DM.</li> <li>Completely missing start or end dates will remain missing, with no imputation applied. Consequently, time to onset and duration of such events will be missing</li> </ul> |
| Concomitant<br>Medications/Medical<br>History | <ul> <li>Partial dates for any concomitant medications recorded in the CRF will be imputed using the following convention: <ul> <li>If the partial date is a start date, a '01' will be used for the day and 'Jan' will be used for the month</li> <li>If the partial date is a stop date, a '28/29/30/31' will be used for the day (dependent on the month and year) and 'Dec' will be used for the month.</li> </ul> </li> <li>The recorded partial date will be displayed in listings.</li> </ul> |

# 10.8. Appendix 8: Values of Potential Clinical Importance

## 10.8.1. Laboratory Values

| Haematology | | | | |
|---|---|---|---|---|
| Laboratory Parameter | Units | Category | Clinical Concern Range | |
| | | | Low Flag (< x) | High Flag (>x) |
| | Ratio of | | | |
| Hematocrit | Ratio of | Female | 0.3 | 0.54 |
| | ı | $\Delta$ from BL | | |
| | a/I | | | |
| Haemoglobin | g/L | Female | 80 | 180 |
| | | $\Delta$ from BL | | |
| Lymphocytes | x10 <sup>9</sup> / L | | 8.0 | |
| Neutrophil Count | x10 <sup>9</sup> / L | | 1.5 | |
| Platelet Count | x10 <sup>9</sup> / L | | 100 | 550 |
| While Blood Cell Count (WBC) | x10 <sup>9</sup> / L | | 3 | 22 |

| Liver Function | | | |
|--------------------|--------|----------|------------------------|
| Test Analyte | Units | Category | Clinical Concern Range |
| ALT/SGPT | U/L | High | ≥ 3x ULN |
| AST/SGOT | U/L | High | ≥ 3x ULN |
| AlkPhos | U/L | High | ≥ 3x ULN |
| T Bilirubin | μmol/L | High | ≥ 1.5xULN |
| | μmol/L | | 1.5xULN T. Bilirubin |
| T. Bilirubin + ALT | U/L | High | + |
| | U/L | | ≥ 2x ULN ALT |

## 10.8.2. Vital Signs

| Vital Sign Parameter | Units | Clinical Concern Range | |
|--------------------------|-------|------------------------|-------|
| (Absolute) | | Lower | Upper |
| Systolic Blood Pressure | mmHg | < 85 | > 160 |
| Diastolic Blood Pressure | mmHg | < 45 | > 100 |
| Heart Rate | bpm | < 40 | > 110 |

# 10.9. Appendix 9: Abbreviations & Trade Marks

## 10.9.1. Abbreviations

| Abbreviation | Description |
|---|---|
| AE | Adverse Event |
| AIC | Akaike's Information Criteria |
| A&R | Analysis and Reporting |
| CI | Confidence Interval |
| CPMS | Clinical Pharmacology Modelling & Simulation |
| COC | Combined Oral Contraceptive |
| non-COC | non-Combined Oral Contraceptive |
| CPSSO | Clinical Pharmacology Science & Study Operations |
| CS | Clinical Statistics |
| CSR | Clinical Study Report |
| CTR | Clinical Trial Register |
| CV <sub>b</sub> / CV <sub>w</sub> | Coefficient of Variation (Between) / Coefficient of Variation (Within) |
| DBF | Database Freeze |
| DBR | Database Release |
| DOB | Date of Birth |
| DP | Decimal Places |
| eCRF | Electronic Case Record Form |
| ECG | Electrocardiogram |
| EMA | European Medicines Agency |
| F | Inhaled Bioavailability |
| FDA | Food and Drug Administration |
| FDAAA | Food and Drug Administration Clinical Results Disclosure Requirements |
| FEV1.0 | Forced expiratory volume at 1 minute |
| FPD | Future Pipelines Discovery |
| GSK | GlaxoSmithKline |
| IA | Interim Analysis |
| ICH | International Conference on Harmonization |
| IDMC | Independent Data Monitoring Committee |
| IDSL | Integrated Data Standards Library |
| IH | Inhaled |
| IM | Intramuscular |
| IMMS | International Modules Management System |
| IP | Investigational Product |
| I.U. | International units |
| IV | Intravenous |
| MMRM | Mixed Model Repeated Measures |
| PCI | Potential Clinical Importance |
| PCPS | Projects, Clinical Platforms and Sciences |
| PD | Pharmacodynamic |
| PDMP | Protocol Deviation Management Plan |
| PK | Pharmacokinetic |

| Abbreviation | Description |
|--------------|--------------------------------------------------|
| PP | Per Protocol |
| PopPK | Population PK |
| QC | Quality Control |
| QTcF | Frederica's QT Interval Corrected for Heart Rate |
| QTcB | Bazett's QT Interval Corrected for Heart Rate |
| RAP | Reporting & Analysis Plan |
| SAC | Statistical Analysis Complete |
| SAE | Serious Adverse Event |
| SPDS | Statistics, Programming and Data Sciences |
| SOP | Standard Operation Procedure |
| TA | Therapeutic Area |
| TFL | Tables, Figures & Listings |
| TSL | Third stage of labour |

## 10.9.2. Trademarks

| Trademarks of the GlaxoSmithKline<br>Group of Companies |
|---------------------------------------------------------|
| ROTAHALER |

| Trademarks not owned by the GlaxoSmithKline Group of Companies |
|----------------------------------------------------------------|
| WinNonlin |
# 10.10. Appendix 10: List of Data Displays

# 10.10.1. Data Display Numbering

All displays (Tables, Figures & Listings) will use the term 'Subjects'. The following numbering will be applied for RAP generated displays:

| Section | Tables | Figures |
|------------------|-----------|---------|
| Study Population | 1.7-1.12 | N/A |
| Pharmacokinetic | 2.6-2.8 | 2.8 |
| Safety | 3.17-3.28 | 3.1 |
| Section | List | ings |
| ICH Listings | 35 | -50 |
| Other Listings | 51- | -53 |

# 10.10.2. Mock Example Shell Referencing

Non IDSL specifications will be referenced as indicated and if required example mock-up displays provided in Appendix 11: Example Mock Shells for Data Displays.

| Section | Figure | Table | Listing |
|-----------------|---------|---------|---------|
| Safety | SAFE_FN | SAFE_TN | SAFE_LN |
| Pharmacokinetic | N/A | PK_TN | NA |

### NOTES:

Non-Standard displays are indicated in the 'IDSL / Example Shell' or 'Programming Notes' column as '[Non-Standard] + Reference.'

# 10.10.3. Deliverables

| Delivery [Priority] [1] | Description |
|---|---|
| DR [1] | Prior to DBR. Dry Run for Study Pop, Safety displays |
| SAC | Final Statistical Analysis Complete |

### NOTES:

<sup>1.</sup> Indicates priority (i.e. order) in which displays will be generated for the reporting effort

# 10.10.4. Study Population Tables

| Study | Study Population Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| Subjec | t Disposition | | | | |
| 1.7. | Safety | ES1 | Summary of Subject Disposition for the Subject Conclusion Record | ICH E3, FDAAA, EudraCT | DR [1], SAC |
| 1.8. | Enrolled | NS1 | Summary of Number of Subjects Enrolled by Country and Site ID | EudraCT/Clinical Operations | DR [1], SAC |
| Popula | tion Analysed | | | | |
| 1.9. | Screened | SP1 | Summary of Study Populations | | DR [1], SAC |
| Demog | Demographic and Baseline Characteristics | | | | |
| 1.10. | Safety | DM1 | Summary of Demographic Characteristics | ICH E3, FDAAA, EudraCT | DR [1], SAC |
| 1.11. | Enrolled | DM11 | Summary of Age Ranges | EudraCT | DR [1], SAC |
| 1.12. | Safety | DM5 | Summary of Race and Racial Combinations | ICH E3, FDA, FDAAA, EudraCT | DR [1], SAC |

# 10.10.5. Pharmacokinetic Tables

| Pharmacol | Pharmacokinetic Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| PK Concer | ntration Data | | | | |
| 2.6. | PK | pkct1 | Summary of Plasma Concentration-time Data | Page by subjects before study restart, subjects after restart and all subjects together. | SAC |
| 2.7. | PK | PK_T1 | Summary of Derived Plasma Pharmacokinetic Parameters (untransformed data) | Page by subjects before study restart, subjects after restart and all subjects together. This will be an overall summary and will not be displayed by timepoints. | SAC |
| 2.8. | PK | PK_T2 | Summary of Number and Percentage of Subjects with Measurable Concentrations | Page by subjects before study restart, subjects after restart and all subjects together. This will be an overall summary and will not be displayed by timepoints. | SAC |

# 10.10.6. Pharmacokinetic Figures

| Pharmacokinetic | Pharmacokinetic Figures | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example<br>Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| Individual Conce | ntration Plots | | | | |
| 2.8. | PK | pkcf6 | Individual Subject Plasma Concentration-time Plot (Linear and Semi-log) by Treatment | By Treatment, Page by subjects before study restart, subjects after restart and all subjects together | SAC |

# 10.10.7. Safety Tables

| Safety: Table | Safety: Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example<br>Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| Adverse Eve | ents (AEs) | | | | |
| 3.17. | Safety | AE1 | Summary of All Adverse Events by System Organ Class and Preferred Term | | DR [1], SAC |
| 3.18. | Safety | AE1 | Summary of Drug-Related Adverse Events | | DR [1], SAC |
| 3.19. | Safety | AE1 | Summary of Non-Serious Adverse Events | | DR [1], SAC |
| 3.20. | Safety | AE15 | Summary of Common (>1 Subject) Non-serious Adverse<br>Events by System Organ Class and Preferred Term (Number of<br>Subjects and Occurrences) | FDAAA, EudraCT | DR [1], SAC |
| Serious and | Other Signific | ant Adverse Eve | ents | | |
| 3.21. | Safety | AE16 | Summary of Serious Adverse Events by System Organ Class and Preferred Term (Number of Subjects and Occurrences) | FDAAA, EudraCT | DR [1], SAC |
| 3.22. | Safety | AE1 | Summary of Adverse Events Leading to Permanent Discontinuation of Study Drug or Withdrawal from Study | | DR [1], SAC |

| Safety: Table | Safety: Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example<br>Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| Laboratory: | Laboratory: Hematology | | | | |
| 3.23. | Safety | LB1 | Summary of Haematology Values | | DR [1], SAC |
| 3.24. | Safety | LB1 | Summary of Haematology Changes from Baseline | | DR [1], SAC |
| Vital Signs | | | | | |
| 3.25. | Safety | VS1 | Summary of Vital Signs | | DR [1], SAC |
| 3.26. | Safety | VS1 | Summary of Change from Baseline for Vital Signs | | DR [1], SAC |
| 3.27. | Safety | VS7 | Summary of Vital Sign Results Relative to Potential Clinical Importance (PCI) Criteria Post-Baseline Relative to Baseline | | DR [1], SAC |
| Exploratory | Exploratory : Questionnaire Results | | | | |
| 3.28. | Safety | SAFE_T1 | Summary of Device Acceptability Questionnaire for Rotahaler Inhaler | | DR[1], SAC |

# 10.10.8. Safety Figure

| Safety: | Safety: Figures | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| Adverse | Adverse Events | | | | |
| 3.1. | Safety | LB10 | Safety Summary Plot of Pre and Post-Delivery Haemaglobin | IDSL Include the timepoints in the x-axis and values in the y-axis | DR[1], SAC |

# 10.10.9. ICH Listings

| ICH: Listings | | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| Subject | Disposition | | | | <u>.</u> |
| 35 | Screened | ES7 | Listing of Reasons for Screening Failure | | DR [1], SAC |
| 36. | Safety | ES2 | Listing of Reasons for Withdrawal | | DR [1], SAC |
| 37. | Safety | TA1 | Listing of Randomised and Actual Treatments | | DR [1], SAC |
| Protoco | l Deviations | | | • | • |
| 38. | Safety | DV2 | Listing of Important Protocol Deviations | | DR [1], SAC |
| 39. | Safety | IE3 | Listing of Participants with Inclusion/Exclusion Criteria Deviations | | DR [1], SAC |
| Populat | ions Analysed | | | | |
| 40. | Enrolled | SP3 | Listing of Participants Excluded from Analysis Population | | DR [1], SAC |
| Demogr | aphic and Bas | eline Characteris | tics | | <u> </u> |
| 41. | Safety | DM2 | Listing of Demographic Characteristics | | DR [1], SAC |
| 42. | Safety | DM9 | Listing of Race | | DR [1], SAC |
| Prior an | d Concomitan | t Medications | | | |
| 43. | Safety | CM3 | Listing of Concomitant Medications | | DR [1], SAC |
| Exposure and Treatment Compliance | | | | | |
| 44. | Safety | EX3 | Listing of Exposure Data | | DR [1], SAC |
| Adverse | Adverse Events | | | | |
| 45. | Safety | AE8 | Listing of All Adverse Events | | DR [1], SAC |
| 46. | Safety | AE7 | Listing of Subject Numbers for Individual Adverse Events | | DR [1], SAC |

| ICH: Lis | ICH: Listings | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| Serious | Serious and Other Significant Adverse Events | | | | |
| 47. | Safety | AE8 | Listing of Serious Adverse Events | | DR [1], SAC |
| 48. | Safety | AE8 | Listing of Adverse Events Leading to Withdrawal from Study | | DR [1], SAC |
| All Lab | oratory | | | | |
| 49. | Safety | LB5 | Listing of All Hematology Data | All PCI criteria will be flagged | DR [1], SAC |
| Vital Si | Vital Signs | | | | |
| 50. | Safety | VS4 | Listing of All Vital Signs Data | All PCI criteria will be flagged | DR [1], SAC |

# 10.10.10. Non-ICH Listings

| Non-IC | Non-ICH: Listings | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| Safety | | | | | |
| 51. | Safety | SAFE_L1 | Listing of Device Acceptability Questionnaire for Rotahaler Inhaler | | DR [1], SAC |
| PK Con | centration | | | | |
| 52. | PK | PK07 | Listing of Plasma Pharmacokinetic Concentration-Time Data | | SAC |
| 53. | PK | PK13 | Listing of Derived Plasma Pharmacokinetic Parameters | | SAC |

# 10.11. Appendix 11: Mock Shell

Example: SAFE\_T1
Protocol: 205920 Page 1 of 2

Population: Safety

Table x.xx

Summary of Device Acceptability Questionnaire for Rotahaler Inhaler

| | Total<br>(N=XX) |
|--------------------------------------|-----------------|
| Feel Confident Received the Medicine | |
| n | XX |
| Yes | xx (xx%) |
| No | xx (xx%) |
| Neutral | xx (xx%) |
| Decline to Answer | xx (xx%) |
| Find This Inhaler Easy to Use | |
| n | XX |
| Yes | xx (xx%) |
| No | xx (xx%) |
| Neutral | xx (xx%) |
| Decline to Answer | xx (xx%) |
| Prefer Inhaler Instead of Injection | |
| n | XX |
| Yes | xx (xx%) |
| No | xx (xx%) |
| Neutral | xx (xx%) |
| Decline to Answer | xx (xx%) |

2019N402257\_00 205920

Example: SAFE\_T1
Protocol: 205920
Population: Safety

Page 2 of 2

Table x.xx

Summary of Device Acceptability Questionnaire for Rotahaler Inhaler

Total (N=XX)

\_\_\_\_\_

This Inhaler Acceptable to Administer

# 2019N402257\_00 205920

Page 1 of n

Example : SAFE\_L1
Protocol : GR121619 Population : Safety

Listing SAFE\_T1
Listing of Device Acceptability Questionnaire for Rotahaler Inhaler

| Site Id<br>Subj Id | · | Date | Question | Response |
|---|---|---|---|---|
| Xxxx/PPD | PERIOD 1 GRP1 | PPD | Feel Confident Received the Medicine<br>Find This Inhaler Easy to Use<br>Prefer Inhaler Instead of Injection<br>This Inhaler Acceptable to Administer | Yes<br>Yes<br>Yes<br>Yes |
| Xxxx/PPD | PERIOD 1 GRP1 | PPD | Feel Confident Received the Medicine<br>Find This Inhaler Easy to Use<br>Prefer Inhaler Instead of Injection<br>This Inhaler Acceptable to Administer | Neutral<br>Yes<br>Yes<br>Yes |

Page 1 of xx

### **CONFIDENTIAL**

Example: PK\_T1

Population: Pharmacokinetic {Group}

Table x.x
Summary of Derived [Analyte] [Matrix] Pharmacokinetic Parameters {by Group}

| Parameter | Treatment | Ν | n | n* | Median | Range |
|---|---|---|---|---|---|---|
| AUC(0-t) (units) | 400mcg | 24 | 24<br>24 | XXXX.XX<br>XXXX.XX | NC<br>xxxx.xx | NC to NC<br>NC to xx |
| | 17mg | 24 | 24<br>23 | XXXX.XX<br>XXXX.XX | XXXX.XX<br>XXXX.XX | XXXX.X<br>XXXX.X |
| Cmax (units) | 400mcg | 24 | 24<br>23 | XXXX.XX<br>XXXX.XX | XXXX.XX<br>XXXX.XX | XXXX.X<br>XXXX.X |
| | 17mg | 24 | 24<br>21 | XXXX.XX<br>XXXX.XX | xxxx.xx<br>xxxx.xx | XXXX.X<br>XXXX.X |

NC = non calculable due to NQ concentrations

NA = not applicable due to insufficient data to derive summary measure

n = Number of subjects with non-missing observations (including imputed NC values)

 $n^*$  = Number of subjects for whom parameter cannot be derived because of NQ concentrations

Note: for Cmax and AUC, NCs were imputed prior to derivation of summary statistics; No NC values were imputed for tmax.

Cmax imputed with ½ LLQ (5 pg/mL)

AUC(0-t) imputed with ½ lowest observed AUC(0-t) (5.45 pg.h/mL)

Example: PK\_T2
Population: Pharmacokinetic Page 1 of xx

Table x.x Summary of Number and Percentage of Subjects with Measurable Concentrations

| Treatment (mcg) | N | n | Number | of measurable | Concentrations | s in the Concentr | ation-time Profile |
|---|---|---|---|---|---|---|---|
| (mog) | | | 0 | 1 | 2 | 3 | >/=4 but <7 |
| 400 | 8 | 8 | 2(25%) | 2 (25%) | 1 (12.5 %) | 1 (12.5%) | 2 (25%) |
| 17 | 7 | 7 | 5 (71%) | 0 (0%) | 0 (0%) | 0 (0%) | 2 (29%) |

n=Number of subjects with non-missing observations (including NC values)

### The GlaxoSmithKline group of companies

205920

| Division | : | Worldwide Development |
|------------------|---|-----------------------------------|
| Information Type | : | Reporting and Analysis Plan (RAP) |

| Title | : | Reporting and Analysis Plan (for Group 2 reporting) for a randomized, open-label study to characterize the pharmacokinetics of inhaled oxytocin (GR121619) compared with IM oxytocin in women in the third stage of labour, and with IV oxytocin in non-pregnant, non-lactating women of childbearing potential. |
|---|---|---|
| <b>Compound Number</b> | : | GR121619 |
| <b>Effective Date</b> | : | 16-JAN-2019 |

## **Description:**

- The purpose of this RAP is to describe the planned analyses and output to be included in the Clinical Study Report for Protocol 205920.
- This RAP is intended to describe the Group 2 analyses required for the study.
- This RAP will be provided to the study team members to convey the content of the Statistical Analysis Complete (SAC) deliverable for Group 2.

### **RAP Author(s):**

| Approver | Date | Approval Method |
|------------------------------------------|-------------|-----------------|
| Associate Statistician (FPD, SPDS India) | N/A | N/A |
| PPD Statistics Director (FPD, SPDS) | 09-JAN-2019 | e-signature |

Copyright 2019 the GlaxoSmithKline group of companies. All rights reserved. Unauthorised copying or use of this information is prohibited.

## The GlaxoSmithKline group of companies

205920

# **RAP Team Approvals:**

| Approver | Date | Approval Method |
|---|---|---|
| Clinical Development Manager, RD PCPS<br>CPSSO | 09-JAN-2019 | e-signature |
| Head, RD Respiratory HUP 2 | 09-JAN-2019 | e-mail |
| Manager, Clinical Pharmacology, CPMS | 09-JAN-2019 | e-signature |
| Manager Data Management, CPSSO Data Management Respiratory | 09-JAN-2019 | e-signature |
| Medical Director, SERM, CMO GCSP SERM US | 16-JAN-2019 | e-mail |
| Principal Programmer/Analyst, RD PCPS Qsci<br>Clinical Statistics 9B2 | 10-JAN-2019 | e-signature |

# **Clinical Statistics and Clinical Programming Line Approvals:**

| Approver | Date | Approval Method |
|---|---|---|
| Biostatistics and Programming Manager, SPDS India | 09-JAN-2019 | e-signature |
| PPD Programming Manager, RD PCPS Qsci Clinical Statistics 9B | 09-JAN-2019 | e-signature |

205920

## **TABLE OF CONTENTS**

| | | | PAGE |
|---|---|---|---|
| 1. | INTRO | ODUCTION | 5 |
| 2. | SUMN | MARY OF KEY PROTOCOL INFORMATION | 5 |
| ۷. | 2.1. | Changes to the Protocol Defined Statistical Analysis Plan | |
| | 2.2. | Study Objective(s) and Endpoint(s) | 6 |
| | 2.3. | Study Design | |
| | 2.4. | Statistical Hypotheses / Statistical Analyses | |
| 3. | PLAN | NNED ANALYSES: GROUP 2 | 10 |
| | 3.1. | Interim Analyses: Group 2 | 10 |
| | 3.2. | Final Analyses | |
| 4. | ANAL' | YSIS POPULATIONS | 10 |
| | 4.1. | Protocol Deviations | 11 |
| 5. | CONS | SIDERATIONS FOR DATA ANALYSES AND DATA HANDLING | |
| | CONV | VENTIONS | 12 |
| | 5.1. | Study Treatment & Sub-group Display Descriptors: Group 2 | |
| | 5.2. | Baseline Definitions | 12 |
| | 5.3. | Other Considerations for Data Analyses and Data Handling Conventions | 13 |
| 6. | STUD | DY POPULATION ANALYSES : GROUP 2 | |
| | 6.1. | Overview of Planned Study Population Analyses | 14 |
| 7. | | ETY ANALYSES : GROUP 2 | |
| | 7.1. | Adverse Events Analyses | |
| | 7.2. | Clinical Laboratory Analyses | |
| | 7.3. | Other Safety Analyses | 15 |
| 8. | PHAR | RMACOKINETIC ANALYSES : GROUP 2 | 16 |
| | 8.1. | Primary Pharmacokinetic Analyses : Group 2 | 1 <mark>6</mark> |
| | | 8.1.1. Endpoint / Variables : Group 2 | |
| | | 8.1.1.1. Drug Concentration Measures : Group 2 | |
| | | 8.1.1.2. Derived Pharmacokinetic Parameters: Group | |
| | | 8.1.2. Summary Measure: Group 2 | 17 |
| | 0.0 | 8.1.3. Population of Interest : Group 2 | 18 |
| | 8.2. | POPULATION PHARMACOKINETIC (POPPK) ANALYSES | |
| | 8.3. | Exploratory Pharmacokinetic Analyses: Group 2 | |
| | | 8.3.1. Endpoint / Variables : Group 2 | |
| | | 8.3.2. Summary Measure: Group 2 | |
| | | 8.3.4. Statistical Analyses / Methods: Group 2 | |
| | | 8.3.4.1. Statistical Methodology Specification | |
| 9. | RFFF | ERENCES | 21 |
| | | ENDICES | 22 |
| 7() | ハレレト | -NI III -> | .,,, |

| 10.1. | | x 1: Protocol Deviation Management and Definitions for Per Population | 22 |
|---|---|---|---|
| 10.2 | | x 2: Schedule of Activities | |
| 10.2. | 10.2.1. | Protocol Defined Schedule of Events : Group 2 | |
| | 10.2.1. | 10.2.1.1. Time & Events General Overview | |
| | | 10.2.1.2. Time & Events General Overview | |
| 10.3. | Annondi | | |
| 10.3. | | x 3: Assessment Windows | 20 |
| 10.4. | | x 4: Study Phases and Treatment Emergent Adverse | 26 |
| | 10.4.1. | Study Phases | |
| | | 10.4.1.1. Study Phases for Concomitant Medication | |
| | 10.4.2. | Treatment Emergent Flag for Adverse Events | |
| 10.5. | | x 5: Data Display Standards & Handling Conventions | |
| | 10.5.1. | Reporting Process | |
| | 10.5.2. | Reporting Standards | |
| | 10.5.3. | Reporting Standards for Pharmacokinetic | |
| 10.6. | Appendix | x 6: Derived and Transformed Data | |
| | 10.6.1. | General | |
| | 10.6.2. | Study Population | |
| | 10.6.3 | Safety | |
| 10.7. | | x 7: Reporting Standards for Missing Data | |
| | 10.7.1. | Premature Withdrawals | |
| | 10.7.2. | Handling of Missing Data | |
| | | 10.7.2.1. Handling of Missing and Partial Dates | |
| 10.8. | Appendix | x 8: Values of Potential Clinical Importance | 34 |
| | 10.8.1. | Laboratory Values | |
| | 10.8.2. | ECG | |
| | 10.8.3. | Vital Signs | |
| 10.9. | | x 11: Abbreviations & Trade Marks | 36 |
| | 10.9.1. | Abbreviations | |
| | 10.9.2. | Trademarks | 37 |
| 10.10. | Appendix | x 12: List of Data Displays | |
| | | Data Display Numbering | |
| | | Mock Example Shell Referencing | |
| | | Deliverables | |
| | | Study Population Tables | |
| | | Pharmacokinetic Tables | |
| | 10.10.6. | Pharmacokinetic Figures | 41 |
| | | Safety Tables | |
| | | ICH Listings | |
| | | Non-ICH Listings | |
| 10.11. | | x 13: Example Mock Shells for Data Displays | |

205920

### 1. INTRODUCTION

The purpose of this reporting and analysis plan (RAP) is to describe the analyses of Group 2 to be included in the Clinical Study Report for Protocol:

| Revision Chronology: | | |
|---|---|---|
| 2016N281575_00 | 2016-AUG-22 | Original |
| 2016N281575_01 | 2016-OCT-10 | Section 6.2: Inclusion of information on CE marking. |
| 2016N281575_02 | 2018-JAN-04 | Update to PK collection procedures and implementation of instream PK data analysis. Update to location of Secondary Medical Monitor contact |
| | | information. |
| 2016N281575_03 | 30-MAY-2018 | Modification to informal interim and Group 2 analysis plans. |

# 2. SUMMARY OF KEY PROTOCOL INFORMATION

# 2.1. Changes to the Protocol Defined Statistical Analysis Plan

Changes from the originally planned statistical analysis specified in the protocol are outlined in Table 1.

Table 1 Changes to Protocol Defined Analysis Plan

| Protocol | Reporting & Analysis Plan | |
|---|---|---|
| Statistical Analysis Plan | Statistical Analysis Plan | Rationale for Changes |
| To compare the IV pharmacokinetics of oxytocin between Cohort A and Cohort B. | To produce summary<br>statistics for IV Bolus and<br>IV infusion by Cohort | Some participants, received IV Bolus dose and some participants received IV infusion dose. As the number of participants that received IV bolus and IV infusion are too small to allow for a formal stats analysis comparison, summary statistics will be presented instead. |
| All Subjects Population | All Subjects population label changed to Safety population. | To be compliant with the<br>new RAP template |
| Enrolled Population (Defined as all subjects who were enrolled for the trial irrespective of whether they were randomized or not and for whom a record exists on the study database. This population will be used for summarizing screening failure reasons. | All participants who passed screening and entered the study including randomized participants and run in failures Note: Screening failures (who never passed screening even if rescreened) and participants screened but never enrolled into the study (Reserve, Not Used) | To be compliant with the new RAP template |

205920

| Protocol | Reporting & Analysis Plan | Reporting & Analysis Plan |
|---|---|---|
| Statistical Analysis Plan | Statistical Analysis Plan | Rationale for Changes |
| | are excluded from the Enrolled | |
| | population as they did not enter | |
| | the study. | |

# 2.2. Study Objective(s) and Endpoint(s)

Group 1 – Women in Third Stage of Labour (TSL)

| Objectives | ur (TSL) Endpoints |
|---|---|
| Primary Objectives | Primary Endpoints |
| To characterize the pharmacokinetics<br>of single doses of IH oxytocin and 10<br>International Units (I.U.) IM oxytocin in<br>women in TSL. | <ul> <li>Plasma concentration time profile for IH oxytocin and 10 I.U. IM oxytocin.</li> <li>PK parameters: Maximum observed plasma concentration (Cmax), Observed plasma concentrations at 10 minutes (min) postdose (Cp10), Observed plasma concentrations at 20 min post-dose (Cp20), Observed plasma concentrations at 30 min post-dose (Cp30), Time to Cmax (tmax), Area under concentration-time curve (AUC), and Terminal phase half-life (t1/2) will be calculated as data permit.</li> </ul> |
| Secondary Objectives | Secondary Endpoints |
| To evaluate the safety and tolerability of inhaled oxytocin. | General safety parameters: adverse events (AE); absolute values and changes over time of vital signs (blood pressure, heart rate, respiratory rate, temperature). |
| To compare pharmacokinetics of IH oxytocin to 10 I.U. IM oxytocin in women in TSL. | Cmax, Cp10, Cp20, Cp30, Area under the concentration-<br>time curve from time zero (pre-dose) to three hours (h)<br>(AUC[0-3h]) will be compared as data permit. |
| Exploratory Objectives | Exploratory Endpoints |
| Pharmacodynamic effect of IH<br>oxytocin and 10 I.U. IM oxytocin in<br>women in TSL. | Pre and post-delivery haemoglobin |
| <ul> <li>Participant feedback regarding ease<br/>of use, instructions, and perceived<br/>ability of patients to use the<br/>ROTAHALER.</li> </ul> | Questionnaire results from participants. |

Group 2 - Non-pregnant, non-lactating females of child bearing potential

| Objectives | Endpoints |
|---|---|
| Primary Objectives | Primary Endpoints |
| To evaluate the safety and tolerability of IH and IV Oxytocin | <ul> <li>General safety parameters: adverse events; absolute values and changes over time of vital signs (blood pressure, heart rate) and 12-lead electrocardiogram (ECG) parameters (PR, QRS, QT, Corrected QT interval [QTc] intervals) from pre-dose values.</li> <li>Specific respiratory safety parameters: adverse respiratory events as monitored by spirometry including Forced expiratory volume at 1 minute (FEV1.0), respiratory rate, and pulse oximetry.</li> </ul> |
| To characterize the pharmacokinetics | Plasma concentration time profile for IH oxytocin and 5 |

205920

| Objectives | Endpoints |
|---|---|
| of single doses of IH oxytocin and 5 I.U. IV oxytocin. | <ul> <li>I.U. IV oxytocin.</li> <li>PK parameters: Cmax, Cp10, Cp20, Cp30, tmax, AUC, Plasma clearance (CL), volume of distribution and t1/2 will be calculated as data permit.</li> </ul> |
| Exploratory Objectives | Exploratory Endpoints |
| To evaluate endogenous plasma<br>oxytocin concentrations in non-<br>pregnant females in the presence and<br>absence of the combined oral<br>contraceptive. | Pre-dose plasma concentrations of oxytocin. |
| To compare the IH pharmacokinetics of oxytocin between Cohort A (subjects on combined oral contraceptive) and Cohort B (subjects using a non-hormonal form of contraception). | Cp10, Cp20, Cp30, Cmax, AUC(0-3h), Area under the concentration time curve from time zero to infinity (AUC[0-∞]) and t1/2, will be compared as data permit. |
| To compare the IV pharmacokinetics<br>of oxytocin between Cohort A and<br>Cohort B. | Cmax, AUC, t1/2, CL and Volume of distribution (VOD) will be compared as data permit. |

Groups 1 and 2 – Women in TSL and Non-pregnant, non-lactating females of child bearing potential

| Objectives | Endpoints |
|---|---|
| Primary Objectives | Primary Endpoints |
| To compare pharmacokinetics of IH oxytocin between Group 1 and Group 2 | <ul> <li>Cp10, Cp20, Cp30, AUC(0-3h) Cmax, AUC(0-3h)<br/>AUC(0-∞), and t1/2 will be compared as data permit.</li> </ul> |

205920

# 2.3. Study Design



205920

| Overview of S | Overview of Study Design and Key Features |
|---|---|
| | of two dosing sessions: |
| | C: 400 mcg lH oxytocin |
| | D: 5 I.U. IV oxytocin |
| Interim | No formal Interim Analysis are planned, however, PK samples will be analysed and |
| Analysis | preliminary PK parameters derived following completion of approximately 5 women on |
| | each treatment group: 400 mcg IH and 10 I.U. IM to women in TSL (Group 1) and 400 |
| | mcg IH to non-pregnant women on the combined oral contraceptive (Group 2 Cohort |
| | A), in order to assess if dose escalation is required. |

# 2.4. Statistical Hypotheses / Statistical Analyses

No formal hypotheses will be tested, however, the following comparison is of interest:

• Cohort A (inhaled oxytocin) vs Cohort B(inhaled oxytocin)

For each PK endpoint of interest, point estimates and corresponding two-sided 90% confidence intervals will be constructed for the ratio of the geometric mean of the test treatment to the geometric mean of the reference treatment,  $\mu(\text{test})/\mu(\text{reference})$  to provide the range of plausible values for the comparisons of interest.

For IV oxytocin, summary statistics will be produced separately for IV Bolus Oxytocin and IV Infusion Oxytocin. Due to small participant numbers, a formal statistical analysis to compare Cohort A vs Cohort B is not possible for IV Bolus or for IV infusion.

205920

### 3. PLANNED ANALYSES: GROUP 2

## 3.1. Interim Analyses: Group 2

No formal Interim Analysis are planned, however, PK samples will be analysed and preliminary PK parameters derived following completion of approximately 5 women on each treatment group: 400 mcg IH and 10 I.U. IM to women in TSL (Group 1) and 400 mcg IH to non-pregnant women on the combined oral contraceptive (Group 2 Cohort A), in order to assess if dose escalation is required.

# 3.2. Final Analyses

An analysis of Group 2 (non-pregnant volunteers) will be performed once Group 2 has completed to allow for full reporting of non-pregnant volunteer data prior to completion of Group 1.

The final planned primary analyses for Group 2 will be performed after the completion of the following sequential steps:

- 1. All participants in group 2 have completed the study as defined in the protocol
- All required database cleaning activities have been completed for group 2 and final database release (DBR) and database freeze (DBF) for group 2 has been declared by Data Management.
- 3. All criteria for unblinding the randomization codes for group 2 have been met.
- 4. Randomization codes for group 2 have been distributed according to RandAll NG procedures.

### 4. ANALYSIS POPULATIONS

| Population | Definition / Criteria | Analyses Evaluated |
|---|---|---|
| Screened | All participants who were screened for eligibility | <ul> <li>Screen Failures</li> </ul> |
| Enrolled | All participants who passed screening and entered the study including randomized participants and run in failures Note: Screening failures (who never passed screening even if rescreened) and participants screened but never enrolled into the study (Reserve, Not Used) are excluded from the Enrolled population as they did not enter the study. | Study Population |
| Safety | Comprise of subjects who receive at least one dose of study medication. This population will be used for the study population and safety displays. Note: This population will be based on the treatment the participants actually received | <ul><li>Study Population</li><li>Safety</li></ul> |
| Pharmacokinetic<br>(PK) | Subjects in the 'Safety' population for whom a pharmacokinetic sample was obtained and analysed. PK population will be the population for reporting PK data. | • PK |

Refer to Appendix 12: List of Data Displays which details the population used for each display.

205920

### 4.1. Protocol Deviations

Protocol deviations will be tracked by the study team throughout the conduct of the study in accordance with the Protocol Deviation Management Plan.

- o Data will be reviewed prior to freezing the database to ensure all important deviations are captured and categorised on the protocol deviations dataset.
- The SI dataset will include all protocol deviations; the analysis dataset will include only important protocol deviations. The analysis dataset will be used for the listing of important protocol deviations.
- The study endpoints will be reported using the populations detailed in Section 4 of this document regardless of whether the participants deviate from the protocol.
- A separate listing of all inclusion/exclusion criteria deviations will also be provided. This listing will be based on data as recorded on the inclusion/exclusion page of the eCRF.

205920

# 5. CONSIDERATIONS FOR DATA ANALYSES AND DATA HANDLING CONVENTIONS

# 5.1. Study Treatment & Sub-group Display Descriptors: Group 2

| | Treatment Group Descriptions | | |
|---|---|---|---|
| | RandAll NG Data Displays for Reporting | | |
| Code | Description | Description | Order in TLF |
| С | 400 mcg IH oxytocin | 400 mcg IH | 1 |
| D1 | 5 I.U. IV oxytocin | 8.5 mcg IV bolus | 2 |
| D2 | 5 I.U. IV oxytocin | 8.5 mcg IV Infusion | 3 |

Treatment comparisons will be displayed as follows using the descriptors as specified:

### 1. IH Oxytocin (COC) vs IH Oxytocin (non-COC)

If the duration of IV oxytocin dose administered is less than or equal to 2min then the IV dose administered is an IV Bolus dose. If the duration of IV oxytocin dose administered is greater than 2 min then the IV dose administered is an IV Infusion dose. The tables/listings that would display the statistics should display IV oxytocin administered as IV Bolus Oxytocin and IV Infusion Oxytocin. Subjects assigned to treatment code D and received the IV via bolus will be labelled as D1 and those who received IV via infusion will be labelled as D2.

The treatment dosage will be included in the footnotes for the respective tables/listings. If treatment codes have been displayed in the tables/listings the treatment descriptions should be included as footnotes. COC refers to Combined Oral Contraceptive and non-COC refers to non-Combined Oral Contraceptive.

### 5.2. Baseline Definitions

For all endpoints (except as noted in baseline definitions) the baseline value will be the latest pre-dose assessment with a non-missing value. If time is not collected, Day 1 assessments are assumed to be taken prior to first dose and used as baseline.

205920

Baseline definitions for Group 2

| Parameter | Study Assessments Considered as Baseline | | | Baseline Used in |
|---|---|---|---|---|
| | Screening | Day -1 | Day 1 (Pre-Dose) | Data Display |
| Safety | | | | |
| Vital Signs (pressure,<br>heart rate,<br>temperature,<br>respiratory rate) | X | X | X | Day 1 |
| LAB | Х | Х | Х | Day 1 |
| ECG | X | X | X | Day 1 |
| FEV1 | X | X | X | Day 1 |

Unless otherwise stated, if baseline data is missing no derivation will be performed and baseline will be set to missing.

# 5.3. Other Considerations for Data Analyses and Data Handling Conventions

Other considerations for data analyses and data handling conventions are outlined in the appendices:

| Section | Component |
|---------|----------------------------------------------------------------|
| 10.3 | Appendix 3: Assessment Windows |
| 10.4 | Appendix 4: Study Phases and Treatment Emergent Adverse Events |
| 10.5 | Appendix 5: Data Display Standards & Handling Conventions |
| 10.6 | Appendix 6: Derived and Transformed Data |
| 10.7 | Appendix 7: Reporting Standards for Missing Data |
| 10.8 | Appendix 8: Values of Potential Clinical Importance |

205920

### 6. STUDY POPULATION ANALYSES: GROUP 2

# 6.1. Overview of Planned Study Population Analyses

The study population analyses will be based on the Safety & Enrolled population, with screen failures as an exception. The study population displays will be produced page wise, grouped by cohorts A and B

Study population analyses including analyses of subject's disposition, protocol deviations, demographic and baseline characteristics, prior and concomitant medications, and exposure and treatment compliance will be based on GSK Core Data Standards.

Details of the planned displays are provided in Appendix 12: List of Data Displays and will be based on GSK data standards and statistical principles.

205920

### 7. SAFETY ANALYSES: GROUP 2

The safety analyses will be based on the Safety population, unless otherwise specified.

### 7.1. Adverse Events Analyses

Adverse events analyses including the analysis of adverse events (AEs), Serious (SAEs) and other significant AEs will be based on GSK Core Data Standards. The details of the planned displays are provided in Appendix 12: List of Data Displays.

# 7.2. Clinical Laboratory Analyses

Laboratory evaluations including the analyses of Chemistry laboratory tests, Hematology laboratory tests, Urinalysis, and liver function tests will be based on GSK Core Data Standards. The details of the planned displays are in Appendix 12: List of Data Displays.

# 7.3. Other Safety Analyses

The analyses of non-laboratory safety test results including ECGs and vital signs will be based on GSK Core Data Standards, unless otherwise specified. The details of the planned displays are presented in Appendix 12: List of Data Displays.

205920

### 8. PHARMACOKINETIC ANALYSES: GROUP 2

# 8.1. Primary Pharmacokinetic Analyses: Group 2

### 8.1.1. Endpoint / Variables : Group 2

- Plasma concentration time profile for IH oxytocin and 5 I.U. IV oxytocin.
- PK parameters: Cmax, Cp10, Cp20, Cp30, tmax, AUC(including AUC(0-t), AUC(0-inf) and AUC(0-3h)), Plasma clearance (CL), volume of distribution and t1/2 will be calculated as data permit

### 8.1.1.1. Drug Concentration Measures: Group 2

Refer to Appendix 5: Data Display Standards & Handling Conventions (Section 10.5.3. Reporting Standards for Pharmacokinetic)

### 8.1.1.2. Derived Pharmacokinetic Parameters: Group 2

Pharmacokinetic parameters will be calculated by standard non-compartmental analysis according to current working practices and GSK procedures using the currently supported version of WinNonlin. All calculations of non-compartmental parameters will be based on actual sampling times. Pharmacokinetic parameters listed will be determined from the plasma concentration-time data, as data permits.

| Treatment | Parameter | Parameter Description |
|---|---|---|
| IH/IV | Cmax | Maximum observed concentration, determined directly from the concentration-time data. |
| IH/IV | Pre - dose | Quantified concentration in PK sample collected at predose, determined directly from the concentration-time data. |
| IH | Cp10 | Quantified concentration in PK sample collected at 10 minutes (nominal time) post-dose, determined directly from the concentration-time data. |
| IH | Cp20 | Quantified concentration in PK sample collected at 20 minutes (nominal time) post-dose, determined directly from the concentration-time data. |
| IH | Cp30 | Quantified concentration in PK sample collected at 30 minutes (nominal time) post-dose, determined directly from the concentration-time data. |
| IH/IV | tmax | Time to reach Cmax, determined directly from the concentration-time data. |
| IH/IV | AUC(0-t) | Area under the concentration-time curve from time zero to the time of the last quantifiable concentration (C(t)) will be calculated using the linear trapezoidal rule for each incremental trapezoid and the log trapezoidal rule for each decremental trapezoid. |
| IH/IV | AUC (0-inf) | Area under the concentration-time curve extrapolated to infinity will be calculated as: AUC = AUC(0-t) + C(t) / lambda_z |
| IH/IV | AUC(0-3h) | Area under the concentration-time curve from time zero to 3 h post-dose |
| IV | Plasma clearance<br>(CL) | Plasma clearance (a volume per time, i.e. a flow) expresses the overall ability of the body to eliminate a drug by scaling the drug elimination rate (amount per time) by the corresponding plasma concentration level. |

205920

| Treatment | Parameter | Parameter Description |
|---|---|---|
| IV | VOD | Volume of distribution of a drug gives information on its distribution in the body. Calculated as VD=Total amount of blood in the body/Drug blood plasma concentration. |
| IH/IV | t1/2 | Apparent terminal half-life will be calculated as: t½ = ln2 / Lambda_z (NOTE: Lambda_z is the terminal phase rate constant). |
| IH/IV | Clast | Last observed quantifiable concentration |
| IH/IV | tlast | Time of the last observed quantifiable concentration |
| IH/IV | Lambda_z | The first order rate constant associated with the terminal (log-linear) portion of the concentration-time curve. |
| IH/IV | Lambda_z_lower | First time point used in computing Lambda_z. |
| IH/IV | Lambda_z_upper | Last time point used in computing Lambda_z. |
| IH/IV | #pts | Number of points used in computing Lambda_z. |
| IH/IV | r-squared | R-squared of Lambda_z computation. |
| IH/IV | AUC(0-inf)/D | AUC(0-inf) corrected for dose |

#### NOTES:

Additional parameters may be included as required.

The absolute bioavailability (F) will be derived for each subject using the formula outlined below. If dose normalised  $AUC(0-\infty)$  cannot be determined this will be substituted with dose normalised AUC(0-t) for that profile. All PK parameters (including the derived inhaled bioavailability, F) will be listed and summarised.

$$F = \frac{AUC(0-\infty)_{inhaled} / Dose_{inhaled}}{AUC(0-\infty)_{IV} / Dose_{IV}}$$

The conversion factor to normalise IV doses is 1 IU = 1.7 mcg oxytocin

# 8.1.2. Summary Measure: Group 2

Pharmacokinetic data will be presented in graphical and/or tabular form and will be summarized descriptively by IH oxytocin , IV Bolus Oxytocin, IV Infusion Oxytocin for each Cohort (Cohort A and Cohort B). In addition data for the derived absolute bioavailability, F will also be summarised by cohort.

For each of the parameters the following summary statistics will be calculated

- Untransformed Data: N, n, arithmetic mean, 90% confidence interval (CI) for the arithmetic mean, standard deviation (SD), median, minimum, maximum.
- Loge-transformed Data: Geometric mean, 90% CI for the geometric mean, standard deviation (SD) of loge-transformed data and %CVb.

For tmax, and t1/2 the summary statistics specified for untransformed data above will be

205920

generated.

# 8.1.3. Population of Interest : Group 2

The primary pharmacokinetic analyses will be based on the Pharmacokinetic population, unless otherwise specified.

# 8.2. POPULATION PHARMACOKINETIC (POPPK) ANALYSES

PK samples will be analysed periodically throughout the study duration to enable development of a preliminary population PK model. If appropriate, a population PK analysis may also be conducted on the final data. In addition the oxytocin plasma concentration-time data may be merged with historical data and analysed as part of a population PK meta-analysis. The timeline for these analyses will be independent of the analysis described in this RAP. To support this analysis a NONMEM-specific data file will be generated, the specifications of which are provided in POP PK RAP appendix.

# 8.3. Exploratory Pharmacokinetic Analyses: Group 2

## 8.3.1. Endpoint / Variables : Group 2

- Pre-dose plasma concentrations of oxytocin.
- For IH formulation: Cp10, Cp20, Cp30, Cmax, Tmax, AUC(0-3h), Area under the concentration time curve from time zero to infinity (AUC[0-∞]) and t1/2, will be compared as data permit.
- For IV formulation: Cmax, AUC(0-inf), AUC(0-3h), t1/2, CL and Volume of distribution (VOD) will be compared as data permit.

## 8.3.2. Summary Measure: Group 2

Descriptive Statistics will be produced for Pre-dose plasma concentrations of oxytocin. Pharmacokinetic data will be presented in graphical and/or tabular form and will be summarized descriptively by cohort

As the number of subjects required to statistically compare IV Bolus Oxytocin and IV Infusion Oxytocin between Cohort A and Cohort B is not sufficient, only summary statistics will be produced for IV Bolus Oxytocin and IV Infusion oxytocin. The Inhaled oxytocin will be statistically compared between Cohort A and Cohort B as described in Section 8.3.4

### 8.3.3. Population of Interest: Group 2

The exploratory pharmacokinetic analyses will be based on the Pharmacokinetic population, unless otherwise specified

205920

### 8.3.4. Statistical Analyses / Methods: Group 2

Details of the planned displays are provided in Appendix 12: List of Data Displays and will be based on GSK Data Standards and statistical principles.

The following pharmacokinetic statistical analyses will only be performed, if sufficient data is available (i.e. if subjects have well defined plasma profiles). Pharmacokinetic analysis will be the responsibility of the Clinical Pharmacology Modelling and Simulation Department, (CPMS) and Statistical analyses of the pharmacokinetic parameter data will be the responsibility of Clinical Statistics (CS).

To compare the IH pharmacokinetics of oxytocin between Cohort A (subjects on combined oral contraceptive) and Cohort B (subjects using a non-hormonal form of contraception), point estimates and corresponding two-sided 90% confidence intervals will be computed for Cp10, Cp20, Cp30, Cmax, Tmax, AUC(0-3h), Area under the concentration-time curve from time zero to infinity (AUC[0-∞]) and t1/2.

Data will be loge-transformed prior to analysis using a mixed effect model with a fixed effect term for cohort and a random effect term for subject, with the exception of T1/2 and Tmax which will be analysed non-parametrically using Mann Whitney test.

### 8.3.4.1. Statistical Methodology Specification

### **Endpoint / Variables**

• For IH: - Cp10, Cp20, Cp30, AUC(0-3h), Cmax, Area under the concentration time curve from time zero to infinity (AUC[0-∞]) will be compared as data permit.

Note: These endpoints will be log transformed for analysis.

### **Model Specification**

Mixed Effect model will be used to analyze the data.

**Endpoint:** log transformed PK parameter **Fixed effect:** Cohort (COC/Non-COC)

Random effect: Subject

- The Kenward and Roger method for approximating the denominator degrees of freedom and correcting for bias in the estimated variance-covariance of the fixed effects will be used.
- An unstructured covariance structure for the G matrix will be used.
- In the event that this model fails to converge, alternative covariance structures may be considered such as VC or CS.
- Akaike's Information Criteria (AIC) will be used to assist with the selection of covariance structure.

205920

### **Model Checking & Diagnostics**

- For the Mixed Model, model assumptions will be checked, and appropriate adjustments may be applied based on the data.
- Distributional assumptions underlying the model used for analysis will be examined by
  obtaining a normal probability plot of the residuals and a plot of the residuals versus the fitted
  values (i.e. checking the normality assumption and constant variance assumption of the model
  respectively) to gain confidence that the model assumptions are reasonable.
- If there are any departures from the distributional assumptions, alternative transformations, such as data squared or square root of data, will be explored.
- Non-parametric analyses will be conducted if the normality assumption does not hold.

### **Model Results Presentation**

 Point estimates and corresponding two-sided 90% confidence intervals for the comparison of interest that is Cohort A (COC) vs Cohort B (non-COC) for IH Oxytocin. These will then be back-transformed to provide point estimates and corresponding 90% confidence intervals for the geometric mean ratios (COC/Non-COC)

### **Endpoint / Variables**

• t1/2, Tmax

Note: This endpoint will not be log transformed for analysis

### **Model Specification**

- Mann-Whitney test
- The test will be performed for IH oxytocin only

### **Model Results Presentation**

• Point estimate and 90% confidence interval for the median difference COC-non COC

205920

## 9. REFERENCES

GlaxoSmithKline Document Number 2016N281575\_03 (amendment no.3 – 30-May-2018): A randomized, open-label study to characterize the pharmacokinetics of IH oxytocin (GR121619) compared with IM oxytocin in women in the third stage of labour, and with IV oxytocin in non-pregnant, non-lactating women of childbearing potential.

205920

# 10. APPENDICES

# 10.1. Appendix 1: Protocol Deviation Management and Definitions for Per Protocol Population

This section is not applicable as Per Protocol Population is not defined for this study.
205920

# 10.2. Appendix 2: Schedule of Activities

# 10.2.1. Protocol Defined Schedule of Events: Group 2

### 10.2.1.1. Time & Events General Overview

### Group 2

| | | Study Day | |
|---|---|---|---|
| Procedure | Screening <sup>5</sup> | Main Phase | Follow - Up (7-21<br>days post<br>dose) |
| Informed Consent and Demography | Χ | | |
| Brief Physical Examination | X | X | |
| Medical history | X | | |
| Pregnancy test | Х | X | |
| Alcohol Breath Test, Smokerlyzer, Urine Drug Screen <sup>1</sup> | χ | X | |
| HIV, Hep B and Hep C screen <sup>2</sup> | X | | |
| Inhaler device training / education session | χ | | |
| Laboratory assessments (including liver chemistries) | X | X | |
| Immunogenicity sample | 9 | X | X |
| 12-lead ECG | X <sup>4</sup> | X | |
| CardiacTelemetry | | Х | |
| Vital signs <sup>3</sup> | X | X | |
| Spirometry (FEV-1) <sup>4</sup> | Χ | Х | |
| Admission to unit | | X | |
| Pharmacokinetic blood sample | Х | Х | |
| Oxytocin Administration (IH or IV) | | X | |
| Prior / concomitant medication review | Х | Х | X |
| AE review | | continuous review | |
| SAE review | | continuous revie | w |
| Discharge from unit | | X | |

- 1. Smokerlyzer at PI/designee discretion if smoking history in question.
- 2. If test otherwise performed within 3 months prior to first dose of study treatment, repeat testing at screening is not required.
- 3. Includes blood pressure, heart rate, temperature, respiratory rate, and SpO2.
- 4. Performed in triplicate.
- 5. To be completed within 28 days of randomization.

205920

#### 10.2.1.2. Time & Events - Main Phase Procedures

Group 2 - Sessions 1 and 2

| | | Time | Post Dos | se | | | | | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Procedure | Pre-<br>dose | 2<br>min | 3<br>min | 5<br>min | 8<br>min | 10<br>min | 15<br>min | 20<br>min | 30<br>min | 45<br>min | 1 hr | 1.5 hr | 2 hr | 2.5 hr | 3 hr | 4 hr |
| Brief Physical Exam | X | | | | | | | | | | | | | | | |
| Pregnancy Test | Χ | | | | | | | | | | | | | | | |
| Alcohol Breath Test, Smokerlyzer, Urine<br>Drug Screen <sup>1</sup> | χ | | | | | | | | | | | | | | | |
| Vital signs <sup>2</sup> | X | | | χ | | | χ | | X | | χ | | | | | X |
| 12-lead ECG | Χ | χ | | | | χ | | X | X | | χ | | | | | χ |
| CardiacTelemetry | - | | | | C | ntinuou | } | | | | - | | | | | |
| Spirometry <sup>3</sup> | Χ | | | | | | | | | | X | | | | | |
| Pharmacokinetic blood sample | X5 | χ | χ | X | χ | χ | χ | X | X | χ | χ | χ | X | χ | χ | X |
| Immunogenicity Sample | Χ | | | | | | | | | | | | | | | |
| Laboratory assessments (including liver chemistries) | χ | | | | | | | | | | | | | | | X |
| Prior medication review | X | | | | | | | | | | | | | | | |
| Concomitant medication review | | confinuous review | | | | | | | | | | | | | | |
| AE review | | | | | | | | | continu | ous revie | w | | | | | |
| SAE Review | | continuous review | | | | | | | | | | | | | | |
| Discharge from unit <sup>4</sup> | | | | | | | | | | | | | | | | χ |

- 1. Smokerlyzer at Principal Investigator (PI)/designee discretion if smoking history in question.
- 2. Includes blood pressure, heart rate, temperature, respiratory rate, and SpO2
- 3. FEV 1.0 will be performed in triplicate at each time point. Record all three values on source document, and record best effort in eCRF.
- 4. Discharge at PI discretion, no sooner than 4-hours post-dose.
- 5. 3 pre-dose samples: approximately 1 hr pre-dose, 30 minutes pre-dose, and 15 minutes pre-dose

205920

# 10.3. Appendix 3: Assessment Windows

No assessment windows will be applied.

205920

# 10.4. Appendix 4: Study Phases and Treatment Emergent Adverse Events

# 10.4.1. Study Phases

Assessments and events will be classified according to the time of occurrence relative to study treatment.

| Study Phase | Definition |
|---|---|
| Pre-Treatment | Date ≤ Study Treatment Start Date |
| On-Treatment | Study Treatment Start Date ≤ Date ≤ Study Treatment Stop Date |
| Post-Treatment | Date > Study Treatment Stop Date |

### 10.4.1.1. Study Phases for Concomitant Medication

| Study Phase | Definition |
|---|---|
| Prior | If medication end date is not missing and is before 28 days prior to screening visit |
| Concomitant | Any medication that is not a prior |

### NOTES:

 Please refer to Appendix 7: Reporting Standards for Missing Data for handling of missing and partial dates for concomitant medication. Use the rules in this table if concomitant medication date is completely missing.

205920

# 10.4.2. Treatment Emergent Flag for Adverse Events

| Flag | Definition |
|---|---|
| Treatment<br>Emergent | <ul> <li>Any AE's occurring after Period 1 dosing and before Period 2 dosing (predose),<br/>will be considered as Period 1 AE's. Any AE's occurring after Period 2 dosing will<br/>be considered as Period 2 AE's.</li> </ul> |
| | <ul> <li>For studies with greater than one treatment period (e.g., crossover study), if AE onset is during one period and worsens during a later period it would be counted in both periods.</li> </ul> |

### NOTES:

- If the study treatment stop date is missing, then the AE will be considered to be On-Treatment.
- Time of study treatment dosing and start/stop time of AEs should be considered, if collected.

205920

# 10.5. Appendix 5: Data Display Standards & Handling Conventions

### 10.5.1. Reporting Process

| Software | |
|---|---|
| The currently supply | The currently supported versions of SAS software 9.4 will be used. |
| Reporting Area | |
| HARP Server | : UK1SALX00175 |
| HARP Compound | : /arenv/arprod/gr121619/mid205920/final_01 |
| Analysis Datasets | Analysis Datasets |
| Analysis datasets | Analysis datasets will be created according to Legacy GSK A&R dataset |
| Generation of RTF Files | |
| RTF files will be generated for summary tables | |

### 10.5.2. Reporting Standards

#### General

- The current GSK Integrated Data Standards Library (IDSL) will be applied for reporting, unless otherwise stated (IDSL Standards Location: https://spope.gsk.com/sites/IDSLLibrary/SitePages/Home.aspx):
  - 4.03 to 4.23: General Principles
  - 5.01 to 5.08: Principles Related to Data Listings
  - 6.01 to 6.11: Principles Related to Summary Tables
  - 7.01 to 7.13: Principles Related to Graphics

#### **Formats**

- All data will be reported according to the actual treatment the subject received unless otherwise stated.
- GSK IDSL Statistical Principles (5.03 & 6.06.3) for decimal places (DP's) will be adopted for reporting of data based on the raw data collected, unless otherwise stated.
- Numeric data will be reported at the precision collected on the eCRF.
- The reported precision from non eCRF sources will follow the IDSL statistical principles but may be adjusted to a clinically interpretable number of DP's.

#### **Planned and Actual Time**

- Reporting for tables, figures and formal statistical analyses:
  - Planned time relative to dosing will be used in figures, summaries, statistical analyses and calculation of any derived parameters, unless otherwise stated.
  - The impact of any major deviation from the planned assessment times and/or scheduled visit days on the analyses and interpretation of the results will be assessed as appropriate.
- Reporting for Data Listings:
  - Planned and actual time relative to study drug dosing will be shown in listings (Refer to IDSL Statistical Principle 5.05.1).
  - Unscheduled or unplanned readings will be presented within the subject's listings.

#### **Unscheduled Visits**

- Unscheduled visits will not be included in summary tables and/or figures.
- All unscheduled visits will be included in listings.

205920

| <b>Descriptive Summary</b> | Statistics | | |
|---|---|---|---|
| Continuous Data | Refer to IDSL Statistical Principle 6.06.1 | | |
| Categorical Data | N, n, frequency, % | | |
| Reporting of Pharmacokinetic Concentration Data | | | |
| Descriptive Summary Statistics | Refer to IDSL Statistical Principle 6.06.1 Assign zero to NQ values (Refer to GUI_51487 for further details) | | |
| Reporting of Pharmac | Reporting of Pharmacokinetic Parameters | | |
| Descriptive Summary<br>Statistics.<br>(Loge Transformed) | Statistics. logged data and between geometric coefficient of variation (CVb (%)) will be | | |
| Parameters Not<br>Being Loge<br>Transformed | Tmax, and t1/2 | | |
| Summary Tables | The following PK parameters will not be summarised: tlast, Lambda_z, Lambda_z_lower, Lambda_z_upper, #pts and r-squared. The following PK parameters will not be log-transformed: Tmax. t1/2 All other parameters will be summarised as log-transformed and non-log-transformed data as described in Section 8.1.2. | | |
| Listings | Include PK Parameters Cmax, Clast, tmax, tlast, AUC(0-3h), AUC(0-t), AUC (0-∞) ),Cp(10), Cp(20), Cp(30) , t1/2, Clearance (IV only), Volume of distribution (IV only), F (Inhaled Bioavailability) Lambda_z, Lambda_z_lower, Lambda_z_upper, #pts and r-squared as data permit | | |
| Reporting of Partial D | lose / No treatment | | |
| | subject has received partial dose or<br>they will be handled as given below: | a subject has received no | treatment in a |
| | Enrolled, Screened Population Safety, PK | | |
| Listings, individual PK figures, Study Population tables uithout period treatment information Include | | | |
| Summary PK figures, Safety and PK tables with treatment information Include Exclude | | | |
| <b>Graphical Displays</b> | | | |
| Refer to IDSL Statistica | al Principals 7.01 to 7.13. | | |

205920

# 10.5.3. Reporting Standards for Pharmacokinetic

| Pharmacokinetic Con | Pharmacokinetic Concentration Data |
|---|---|
| PC Windows Non-<br>Linear (WNL) File | PC WNL file (CSV format) for the non compartmental analysis by Clinical Pharmacology Modelling and Simulation function will be created according to IDSL Standards. Note: Concentration values will be imputed as per GUI_51487 |
| Descriptive Summary<br>Statistics, Graphical<br>Displays and Listings | Refer to IDSL PK Display Standards. Refer to IDSL Statistical Principle 6.06.1. Note: Concentration values will be imputed as per GUI_51487 for descriptive summary statistics/analysis and summarized graphical displays only. |
| NONMEM/Pop PK<br>File | Pop-PK file (CSV format) for the POP-PK analysis by Clinical Pharmacology Modelling and Simulation function will be created according to the data specification detailed in Section 9.1 Data Specification of the Pop-PK RAP (RAP-IVF116828-201558-205920-PopPK, located in Cabinets/Study File/GR121619/_Project/Meta Analysis/ RAP-IVF116828-201558-205920-PopPK) |
| Pharmacokinetic Para | ameter Derivation |
| PK Parameter to be<br>Derived by<br>Programmer | The following PK parameters will be derived by the Programmer: Cp10, Cp20 and Cp30 and pre-dose |
| Pharmacokinetic Para | ameter Data |
| Is NQ impacted PK<br>Parameters Rule<br>Being Followed | Yes, refer to Standards for Handling NQ Impacted PK Parameters |
| Descriptive Summary<br>Statistics, Graphical<br>Displays and Listings | Refer to IDSL PK Display Standards. Refer to Standards for the Transfer and Reporting of PK Data using HARP |

205920

### 10.6. Appendix 6: Derived and Transformed Data

### 10.6.1. **General**

### Multiple Measurements at One Analysis Time Point

- Mean of the measurements will be calculated and used in any derivation of summary statistics but if listed, all data will be presented.
- Participants having both High and Low values for Normal Ranges at any post-baseline visit for safety parameters will be counted in both the High and Low categories of "Any visit post-baseline" row of related summary tables. This will also be applicable to relevant Potential Clinical Importance summary tables.

### **Study Day**

- Calculated as the number of days from First Dose Date:
  - Ref Date = Missing → Study Day = Missing
  - Ref Date < First Dose Date → Study Day = Ref Date First Dose Date</li>
  - Ref Data ≥ First Dose Date → Study Day = Ref Date (First Dose Date) + 1

### 10.6.2. Study Population

#### **Demographics**

#### Age

- GSK standard IDSL algorithms will be used for calculating age.
- Randomization date will be used as reference date to calculate age

### **Body Mass Index (BMI)**

Calculated as Weight (kg) / [Height (m)<sup>2</sup>

#### **Extent of Exposure**

• Number of days of exposure to study drug will be calculated based on the formula:

#### Duration of Exposure in Days = Treatment Stop Date - (Treatment Start Date) + 1

- Participants who were randomized but did not report a treatment start date will be categorised as having zero days of exposure.
- The cumulative dose will be based on the formula:

### **Cumulative Dose = Sum of (Number of Days x Total Daily Dose)**

• If there are any treatment breaks during the study, exposure data will be adjusted accordingly.

205920

### 10.6.3 Safety

### **ECG Parameters**

#### **RR Interval**

• IF RR interval (msec) is not provided directly, then RR can be derived as :

[1] If QTcB is machine read & QTcF is not provided, then :

 $RR = [(QT/QTcB)^{2}]^{1000}$ 

[2] If QTcF is machine read and QTcB is not provided, then:

 $RR = [(QT/QTcF)^{4}]*1000$ 

• If ECGs are manually read, the RR value preceding the measurement QT interval should be collected values THEN do not derive.

#### **Corrected QT Intervals**

- When not entered directly in the eCRF, corrected QT intervals using Bazett's (QTcB) and Fredericia's (QTcF) formulas will be calculated, in msec, depending on the availability of other measurements.
- IF RR interval (msec) is provided or calculated then missing QTcB and/or QTcF will be derived as :

$$QTcB = \frac{QT}{\sqrt{\frac{RR}{1000}}}$$

$$QTcF = \frac{QT}{3\sqrt{\frac{RR}{1000}}}$$

205920

# 10.7. Appendix 7: Reporting Standards for Missing Data

# 10.7.1. Premature Withdrawals

| Element | Reporting Detail |
|---|---|
| General | <ul> <li>Subject study completion (i.e. as specified in the protocol) was defined as who has completed all phases of the study including the follow-up visit(s).</li> <li>Withdrawn subjects may be replaced in the study.</li> <li>All available data from participants who were withdrawn from the study will be listed and all available planned data will be included in summary tables and figures, unless otherwise specified.</li> </ul> |

# 10.7.2. Handling of Missing Data

| Element | Reporting Detail |
|---|---|
| General | Missing data occurs when any requested data is not provided, leading to blank fields on<br>the collection instrument: |
| | <ul> <li>These data will be indicated by the use of a "blank" in subject listing displays. Unless all data for a specific visit are missing in which case the data is excluded from the table.</li> <li>Answers such as "Not applicable" and "Not evaluable" are not considered to be missing data and should be displayed as such.</li> </ul> |
| Outliers | Any participants excluded from the summaries and/or statistical analyses will be documented along with the reason for exclusion in the clinical study report. |

# 10.7.2.1. Handling of Missing and Partial Dates

| Element | Reporting Detail |
|---|---|
| General | Partial dates will be displayed as captured in subject listing displays. |
| Adverse Events | <ul> <li>The eCRF does not allow for the possibility of partial dates. The eCRF and the site need to enter the full date or if not known, they would be required to complete an item level comment bubble to specify why the date is unknown. This would also be documented in the Data Quality Release Report by DM.</li> <li>Completely missing start or end dates will remain missing, with no imputation applied. Consequently, time to onset and duration of such events will be missing</li> </ul> |
| Concomitant<br>Medications/Medical<br>History | <ul> <li>Partial dates for any concomitant medications recorded in the CRF will be imputed using the following convention: <ul> <li>If the partial date is a start date, a '01' will be used for the day and 'Jan' will be used for the month</li> <li>If the partial date is a stop date, a '28/29/30/31' will be used for the day (dependent on the month and year) and 'Dec' will be used for the month.</li> </ul> </li> <li>The recorded partial date will be displayed in listings.</li> </ul> |

205920

# 10.8. Appendix 8: Values of Potential Clinical Importance

# 10.8.1. Laboratory Values

| Haematology | | | | |
|---|---|---|---|---|
| Laboratory Parameter | Units | Category | Clinical Concern Range | |
| | | | Low Flag (< x) | High Flag (>x) |
| | D-4:4 | Male | | 0.54 |
| Hematocrit | Ratio of | Female | | 0.54 |
| | ' | $\Delta$ from BL | ↓0.075 | |
| | /1 | Male | | 180 |
| Haemoglobin | g/L | Female | 180 | |
| | | $\Delta$ from BL | ↓25 | |
| Lymphocytes | x109/ L | | 0.8 | |
| Neutrophil Count | x109/ L | | 1.5 | |
| Platelet Count | x109/ L | | 100 | 550 |
| While Blood Cell Count (WBC) | x109/ L | | 3 | 20 |

| Clinical Chemistry | | | | |
|---|---|---|---|---|
| Laboratory Parameter | Units | Category | Clinical Concern Range | |
| | | | Low Flag (< x) | High Flag (>x) |
| Albumin | g/L | | 30 | |
| Calcium | mmol/L | | 2 | 2.75 |
| Creatinine | umol/L | $\Delta$ from BL | | ↑ <b>44.2</b> |
| Glucose | mmol/L | | 3 | 9 |
| Magnesium | mmol/L | | 0.5 | 1.23 |
| Phosphorus | mmol/L | | 0.80 | 1.60 |
| Potassium | mmol/L | | 3 | 5.5 |
| Sodium | mmol/L | | 130 | 150 |
| Total CO2 | mmol/L | | 18.0 | 32.0 |

| Liver Function | | | |
|--------------------|--------|----------|------------------------|
| Test Analyte | Units | Category | Clinical Concern Range |
| ALT/SGPT | U/L | High | ≥ 2x ULN |
| AST/SGOT | U/L | High | ≥ 2x ULN |
| AlkPhos | U/L | High | ≥ 2x ULN |
| T Bilirubin | µmol/L | High | ≥ 1.5xULN |
| | µmol/L | | 1.5xULN T. Bilirubin |
| T. Bilirubin + ALT | U/L | High | + |
| | U/L | | ≥ 2x ULN ALT |

205920

# 10.8.2. ECG

| ECG Parameter | Units | Clinical Concern Range | |
|----------------------------|-------|------------------------|-------|
| | | Lower | Upper |
| Absolute | | | |
| Absolute QTc Interval msec | | > 450 | |
| Absolute PR Interval msec | | < 110 | > 220 |
| Absolute QRS Interval msec | | < 75 | >110 |

# 10.8.3. Vital Signs

| Vital Sign Parameter | Units | Clinical Concern Range | |
|--------------------------|-------|------------------------|-------|
| (Absolute) | | Lower | Upper |
| Systolic Blood Pressure | mmHg | < 85 | > 160 |
| Diastolic Blood Pressure | mmHg | < 45 | > 100 |
| Heart Rate | bpm | < 40 | > 110 |

205920

# 10.9. Appendix 11: Abbreviations & Trade Marks

# 10.9.1. Abbreviations

| Abbreviation | Description |
|---|---|
| AE | Adverse Event |
| AIC | Akaike's Information Criteria |
| A&R | Analysis and Reporting |
| CI | Confidence Interval |
| CPMS | Clinical Pharmacology Modelling & Simulation |
| COC | Combined Oral Contraceptive |
| 000 | Combined Oral Contraceptive |
| non-COC | non-Combined Oral Contraceptive |
| CPSSO | Clinical Pharmacology Science & Study Operations |
| CS | Clinical Statistics |
| CSR | Clinical Study Report |
| CTR | Clinical Trial Register |
| CV <sub>b</sub> / CV <sub>w</sub> | Coefficient of Variation (Between) / Coefficient of Variation (Within) |
| DBF | Database Freeze |
| DBR | Database Release |
| DOB | Date of Birth |
| DP | Decimal Places |
| eCRF | Electronic Case Record Form |
| ECG | Electrocardiogram |
| EMA | European Medicines Agency |
| F | Inhaled Bioavailability |
| FDA | Food and Drug Administration |
| FDAAA | Food and Drug Administration Clinical Results Disclosure Requirements |
| FEV1.0 | Forced expiratory volume at 1 minute |
| FPD | Future Pipelines Discovery |
| GSK | GlaxoSmithKline |
| IA | Interim Analysis |
| ICH | International Conference on Harmonization |
| IDMC | Independent Data Monitoring Committee |
| IDSL | Integrated Data Standards Library |
| IH | Inhaled |
| IM | Intramuscular |
| IMMS | International Modules Management System |
| IP | Investigational Product |
| I.U. | International units |
| IV | Intravenous |
| MMRM | Mixed Model Repeated Measures |
| PCI | Potential Clinical Importance |
| PCPS | Projects, Clinical Platforms and Sciences |
| PD | Pharmacodynamic |
| PDMP | Protocol Deviation Management Plan |

205920

| Abbreviation | Description |
|--------------|--------------------------------------------------|
| PK | Pharmacokinetic |
| PP | Per Protocol |
| PopPK | Population PK |
| QC | Quality Control |
| QTcF | Frederica's QT Interval Corrected for Heart Rate |
| QTcB | Bazett's QT Interval Corrected for Heart Rate |
| RAP | Reporting & Analysis Plan |
| SAC | Statistical Analysis Complete |
| SAE | Serious Adverse Event |
| SPDS | Statistics, Programming and Data Sciences |
| SOP | Standard Operation Procedure |
| TA | Therapeutic Area |
| TFL | Tables, Figures & Listings |
| TSL | Third stage of labour |

# 10.9.2. Trademarks

| Trademarks of the GlaxoSmithKline<br>Group of Companies |
|---------------------------------------------------------|
| ROTAHALER |

Trademarks not owned by the GlaxoSmithKline Group of Companies
WinNonlin

205920

### 10.10. Appendix 12: List of Data Displays

### 10.10.1. Data Display Numbering

All displays (Tables, Figures & Listings) will use the term 'Subjects'. The following numbering will be applied for RAP generated displays:

| Section | Tables Figures | |
|------------------|-----------------------|-----|
| Study Population | 1.1 to 1.6 | N/A |
| Pharmacokinetic | 2.1 to 2.5 2.1 to 2.7 | |
| Safety | 3.1 to 3.16 N/A | |
| Section | Listings | |
| ICH Listings | 1 to 24 | |
| Other Listings | 25 to 29 | |

### 10.10.2. Mock Example Shell Referencing

Non IDSL specifications will be referenced as indicated and if required example mock-up displays provided in Appendix 13: Example Mock Shells for Data Displays.

| Section | Figure | Table | Listing |
|-----------------|--------|-------|---------|
| Pharmacokinetic | N/A | PK_Tn | N/A |

#### NOTES:

Non-Standard displays are indicated in the 'IDSL / Example Shell' or 'Programming Notes' column as '[Non-Standard] + Reference.'

#### 10.10.3. Deliverables

| Delivery [Priority] [1] | Description |
|---|---|
| DR [1] | Prior to DBR. Dry Run for Study Pop, Safety & PK concentration displays |
| | (Summary Table and Mean/Median plots) |
| DR [2] | Post DBF, prior to SAC. Dry Run for displays not part of Dry run [1] |
| SAC | Final Statistical Analysis Complete |

#### NOTES:

1. Indicates priority (i.e. order) in which displays will be generated for the reporting effort

205920

# 10.10.4. Study Population Tables

| Study | Study Population Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| Subjec | t Disposition | | | | |
| 1.1. | Safety | ES1A | Summary of Participant Disposition for the Participant Conclusion Record | By Cohort<br>ICH E3, FDAAA, EudraCT | DR [1], SAC |
| 1.2. | Enrolled | NS1 | Summary of Number of Subjects Enrolled by Country and Site ID | By Cohort<br>EudraCT/Clinical Operations | DR [1], SAC |
| Popula | tion Analysed | | | | |
| 1.3. | Screened | SP1 | Summary of Study Populations | By Cohort | DR [1], SAC |
| Demog | raphic and Base | line Characteristics | 3 | | |
| 1.4. | Safety | DM3 | Summary of Demographic Characteristics | By Cohort<br>ICH E3, FDAAA, EudraCT | DR [1], SAC |
| 1.5. | Enrolled | DM11 | Summary of Age Ranges | By Cohort EudraCT | DR [1], SAC |
| 1.6. | Safety | DM5 | Summary of Race and Racial Combinations | By Cohort<br>ICH E3, FDA, FDAAA, EudraCT | DR [1], SAC |

205920

### 10.10.5. Pharmacokinetic Tables

| Pharma | acokinetic Tabl | es | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| PK Cor | ncentration Dat | a | | | |
| 2.1. | PK | pkct1 | Summary of Plasma Concentration-time Data | By Cohort | DR [1], SAC |
| PK Der | ived Parameter | 's | | | |
| 2.2. | PK | pkpt1 | Summary of Derived Plasma Pharmacokinetic Parameters (untransformed data) | By Cohort | DR [2], SAC |
| 2.3. | PK | pkpt3 | Summary of Derived Plasma Pharmacokinetic Parameters (log-transformed data) | By Cohort | DR [2], SAC |
| Statisti | cal Analysis Ta | bles | | | |
| 2.4. | PK | PK_T1 | Summary of Statistical Analysis of Loge-transformed Pharmacokinetic Parameters (IH Formulation) | For Cp10, Cp20, Cp30, Cmax, AUC(0-3h) and AUC(0-inf) only. Include treatment dosage in the footnote (Refer Section 5.1) | DR [2], SAC |
| 2.5. | PK | PK_T2 | Summary of Statistical Analysis of un-transformed Pharmacokinetic Parameter (IH Formulation) | For t1/2 and Tmax only<br>Include treatment dosage in the<br>footnote (Refer Section 5.1) | DR [2], SAC |

205920

# 10.10.6. Pharmacokinetic Figures

| Pharmacokinetic Figures | | | | | |
|---|---|---|---|---|---|
| No. | Population IDSL / Example Shell | | Title | Programming Notes | Deliverable<br>[Priority] |
| Individu | ual Concentrati | on Plots | | | |
| 2.1. | PK | pkcf1x | Individual Plasma Concentration-time Plot (Linear and Semi-log) by Subject | By Cohort, By Subject | DR [2], SAC |
| 2.2. | PK | pkcf6 | Individual Subject Plasma Concentration-time Plot (Linear and Semi-log) by Treatment | By Cohort, By Treatment | DR [2], SAC |
| Mean/N | ledian Plots | | | | |
| 2.3. | PK | pkcf4 | Arithmetic Mean (±SD) Plasma Concentration-time Plot (Linear and Semi-log) – Cohort Comparison | Use nominal times in X Axis. By treatment. Produce two curves one for COC and one for non-COC. | DR [1], SAC |
| 2.4. | PK | pkcf5 | Median (range) Plasma Concentration-time Plot (Linear and Semi-log) (IH Formulation)— Cohort Comparison | Use nominal times in X Axis, By treatment | DR [1], SAC |
| 2.5. | PK | pkcf4 | Arithmetic Mean (±SD) Plasma Concentration-time Plot (Linear and Semi-log) – Treatment Comparison | Use nominal times in X Axis. By Cohort. Produce three curves. One each for IH, IV Bolus, IV infusion | DR [1], SAC |
| 2.6. | PK | pkcf5 | Median (range) Plasma Concentration-time Plot (Linear and Semi-log) (IH Formulation)— Treatment Comparison | Use nominal times in X Axis, By Cohort | DR [1], SAC |
| Compa | rative plots | | | | |
| 2.7. | PK | pkpf3 | Comparative Plot of Individual Subject Plasma Pharmacokinetic Parameter Versus Treatment | For all PK Parameter page by<br>Treatment sequence;<br>By Cohort | DR [2], SAC |

205920

# 10.10.7. Safety Tables

| Safety: Tables | | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| Advers | e Events (AEs) | | | | |
| 3.1. | Safety | AE1CP | Summary of All Adverse Events by System Organ Class and Preferred Term | By Cohort | DR [1], SAC |
| 3.2. | Safety | AE1CP | Summary of Drug-Related Adverse Events | By Cohort | DR [1], SAC |
| 3.3. | Safety | AE1CP | Summary of Non-Serious Adverse Events | By Cohort | DR [1], SAC |
| 3.4. | Safety | AE15 | Summary of Common (>1 Subject) Non-serious Adverse Events by System Organ Class and Preferred Term (Number of Subjects and Occurrences) | By Cohort<br>FDAAA, EudraCT | DR [1], SAC |
| Serious | and Other Sig | nificant Adverse | Events | | |
| 3.5. | Safety | AE16 | Summary of Serious Adverse Events by System Organ Class and Preferred Term (Number of Subjects and Occurrences) | By Cohort<br>FDAAA, EudraCT | DR [1], SAC |
| 3.6. | Safety | AE1CP | Summary of Adverse Events Leading to Permanent Discontinuation of Study Drug or Withdrawal from Study | By Cohort | DR [1], SAC |
| Labora | tory: Chemistry | ı | | | |
| 3.7. | Safety | LB1 | Summary of Chemistry Laboratory Values | By Cohort | DR [1], SAC |
| 3.8. | Safety | LB1 | Summary of Change from Baseline for Chemistry Laboratory Values | By Cohort | DR [1], SAC |

205920

| Safety: | Safety: Tables | | | | |
|---|---|---|---|---|---|
| No. | Population IDSL / Example Shell | | Title | Programming Notes | Deliverable<br>[Priority] |
| Labora | tory: Hematolo | gy | | | · |
| 3.9. | Safety | LB1 | Summary of Haematology Laboratory Values | By Cohort | DR [1], SAC |
| 3.10. | Safety | LB1 | Summary of Change from Baseline for Haematology Laboratory Values | By Cohort | DR [1], SAC |
| Spirom | etry | | | | · |
| 3.11. | Safety | LB1 | Summary of Spirometry data | By Cohort. | DR [1], SAC |
| ECG | | | | | |
| 3.12. | Safety | EG1 | Summary of ECG Findings | By Cohort | DR [1], SAC |
| 3.13. | Safety | EG2 | Summary of ECG Values | By Cohort | DR [1], SAC |
| Vital Si | gns | | | | |
| 3.14. | Safety | VS1 | Summary of Vital Signs | By Cohort | DR [1], SAC |
| 3.15. | Safety | VS1 | Summary of Change from Baseline for Vital Signs | By Cohort | DR [1], SAC |
| 3.16. | Safety | VS7 | Summary of Vital Sign Results Relative to Potential Clinical Importance (PCI) Criteria Post-Baseline Relative to Baseline | By Cohort | DR [1], SAC |

205920

# 10.10.8. ICH Listings

| ICH: Listings | | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| Subjec | Subject Disposition | | | | |
| 1. | Screened | ES7 | Listing of Reasons for Screening Failures | By Cohort | DR [1], SAC |
| 2. | Safety | ES3 | Listing of Reasons for Withdrawal | By Cohort | DR [1], SAC |
| 3. | Safety | TA2 | Listing of Randomized and Actual Treatments | By Cohort | DR [1], SAC |
| Protoc | ol Deviations | | | · | |
| 4. | Safety | DV2A | Listing of Important Protocol Deviations | By Cohort | DR [1], SAC |
| 5. | Safety | IE4 | Listing of Participants with Inclusion/Exclusion Criteria Deviations | By Cohort | DR [1], SAC |
| Popula | tions Analysed | | | | |
| 6. | Enrolled | SP3A | Listing of Participants Excluded from Analysis Population | By Cohort | DR [1], SAC |
| Demog | raphic and Bas | eline Characteris | tics | | |
| 7. | Safety | DM4 | Listing of Demographic Characteristics | By Cohort | DR [1], SAC |
| 8. | Safety | DM10 | Listing of Race | By Cohort | DR [1], SAC |
| Prior a | nd Concomitan | t Medications | | | |
| 9. | Safety | CM5 | Listing of Concomitant Medications | By Cohort | DR [1], SAC |
| Exposure and Treatment Compliance | | | | | |
| 10. | Safety | EX4 | Listing of Exposure Data | By Cohort | DR [1], SAC |
| Advers | Adverse Events | | | | |
| 11. | Safety | AE9 | Listing of All Adverse Events | By Cohort | DR [1], SAC |

205920

| ICH: Li | stings | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 12. | Safety | AE7 | Listing of Subject Numbers for Individual Adverse Events | By Cohort | DR [1], SAC |
| Serious | and Other Sig | nificant Adverse | Events | | <u> </u> |
| 13. | Safety | AE9 | Listing of Serious Adverse Events | By Cohort | DR [1], SAC |
| 14. | Safety | AE9 | Listing of Adverse Events Leading to Withdrawal from Study | By Cohort | DR [1], SAC |
| All Lab | oratory | | | | · |
| 15. | Safety | LB6 | Listing of Laboratory Values of Potential Clinical Importance | By Cohort | DR [1], SAC |
| 16. | Safety | LB6 | Listing of All Laboratory Data for Subjects with Any Value of Potential Clinical Importance | By Cohort | DR [1], SAC |
| 17. | Safety | LB6 | Listing of Hematology Values of Potential Clinical Importance | By Cohort | DR [1], SAC |
| 18. | Safety | LB6 | Listing of All Hematology Laboratory Data for Subjects with Any Value of Potential Clinical Importance | By Cohort | DR [1], SAC |
| 19. | Safety | UR2B | Listing of Urinalysis Data | By Cohort | DR [1], SAC |
| ECG | | | | | <u> </u> |
| 20. | Safety | Safety EG4 Listing of All ECG Values for Participants with Any Value of Potential Clinical Importance | | By Cohort | DR [1], SAC |
| 21. | Safety | EG4 | Listing of ECG Values of Potential Clinical Importance | By Cohort | DR [1], SAC |
| 22. | Safety | EG6 | Listing of Abnormal ECG Findings | By Cohort | DR [1], SAC |
| Vital Si | gns | | | | |
| 23. | Safety | VS5 | Listing of All Vital Signs Data for Subjects with Any Value of Potential Clinical Importance | By Cohort | DR [1], SAC |
| 24. | Safety | VS5 | Listing of Vital Signs of Potential Clinical Importance | By Cohort | DR [1], SAC |

205920

# 10.10.9. Non-ICH Listings

| Non-ICH: Listings | | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| Safety | | | | | |
| 25. | Safety | EG4 | Listing of Spirometry data | By Cohort | DR [1], SAC |
| PK Cor | centration | | | | |
| 26. | PK | PK08 | By Cohort | DR [2], SAC | |
| PK Para | ameter | | | | |
| 27. | PK | PK14 | Listing of Derived Plasma Pharmacokinetic Parameters | By Cohort | DR [2], SAC |
| 28. | PK | N/A | Raw SAS output for Summary of Statistical Analysis of Loge-<br>transformed Pharmacokinetic Parameters for IH formulation | For Cp10, Cp20, Cp30, Cmax, AUC(0-3h) and AUC(0-inf) only. Include treatment dosage in the footnote (Refer Section 5.1). Include footnotes present in the corresponding analysis table | DR [2], SAC |
| 29. | PK | N/A | Raw SAS output for Summary of Statistical Analysis of untransformed Plasma Pharmacokinetic Parameter for IH formulation | For t/2 and Tmax only Include treatment dosage in the footnote (Refer Section 5.1). Include footnotes present in the corresponding analysis table | DR [2], SAC |

205920

### 10.11. Appendix 13: Example Mock Shells for Data Displays

Example : PK\_T1 Page 1 of n

Protocol : GR121619
Population : Pharmacokinetic

Table PK\_T1
Summary of Statistical Analysis of log transformed GR121619 Pharmacokinetic Parameters for IH formulation

| Parameter (units) | Comparison | Comparison Geo | | Geom.LsMean Ratio | | Ratio | 90%<br>Confidence Interval |
|---|---|---|---|---|---|---|---|
| | | n | Test | n | Ref | | Confidence interval |
| AUC(0-t)(µg.h/mL) | COC vs non-COC | XX | x.xxx | XX X | <br>x.xxx | x.xxx | (x.xxx, x.xxx) |

Note:1. Mixed Effect Model has been used for the analysis. Cohort (COC/Non-COC is fitted as Fixed Effect. Subject is fitted as Random Effect.

<sup>2.</sup> \_\_\_\_\_ covariance structure is used

205920

Example Protocol : PK\_T2 : GR121619 Page 1 of n

Population : Pharmacokinetic

Table PK\_T2 Summary of Statistical Analysis of un-transformed Pharmacokinetic Parameter IH Formulation

| Parameter (units) | Comparison | Median | | | | Diff | 90% |
|---|---|---|---|---|---|---|---|
| | | | | | - | | Confidence Interval |
| | | n | Test | n | Ref | | |
| T1/2 | COC vs non-COC | ×x | x.xxx | xx | x.xxx | x.xxx | (x.xxx, x.xxx) |

Appropriate footnotes to be used